# Journey of Transformation Curriculum for Native American Adolescents (JOT)

# NCT05274217

Teresa Evans-Campbell, PhD

Study Protocol

IRB Approved 03-16-2021



The Human Subjects Division (HSD) strives to ensure that people with disabilities have access to all services and content. If you experience any accessibility-related issues with this form or any aspect of the application process, email <a href="https://hsd.nicolor.nico

# **INSTRUCTIONS**

- This form is only for studies that will be reviewed by the UW IRB. Before completing this form, check HSD's website to confirm that this should not be reviewed by an external (non-UW) IRB.
- <u>If you are requesting a determination</u> about whether the planned activity is human subjects research or qualifies for exempt status, you may skip all questions except those marked with a . For example 1.1 must be answered.
- Answer all questions. If a question is not applicable to the research or if you believe you have already answered a question elsewhere in the application, state "NA" (and if applicable, refer to the question where you provided the information). If you do not answer a question, the IRB does not know whether the question was overlooked or whether it is not applicable. This may result in unnecessary "back and forth" for clarification. Use non-technical language as much as possible.
- To check a box, place an "X" in the box. To fill in a text box, make sure your cursor is within the gray text box bar before typing or pasting text.
- For collaborative or multi-site research, describe only the UW activities unless you are requesting that the UW IRB provide the review and oversight for non-UW collaborators or co-investigators as well.
- You may reference other documents (such as a grant application) if they provide the requested information in non-technical language. Be sure to provide the document name, page(s), and specific sections, and upload it to *Zipline*. Also, describe any changes that may have occurred since the document was written (for example, changes that you've made during or after the grant review process). In some cases, you may need to provide additional details in the answer space as well as referencing a document.

| INDEX | | |
|---|---|---|
| 1 <u>Overview</u> | 6 Children (Minors) and Parental Permission | 10 Risk / Benefit Assessment |
| 2 Participants | 7 Assent of Children (Minors) | 11 Economic Burden to Participants |
| 3 Non-UW Research Setting | 8 Consent of Adults | 12 Resources |
| 4 Recruiting and Screening Participants | 9 Privacy and Confidentiality | 13 Other Approvals, Permissions, and Regulatory Issues |
| 5 Procedures | | |

APPLICATION IRB Protocol

# **1 OVERVIEW**

**Study Title:** 

Journey of Transformation

**1.1**)Home institution. Identify the institution through which the lead researcher listed on the IRB application will conduct the research. Provide any helpful explanatory information.

In general, the home institution is the institution (1) that provides the researcher's paycheck and that considers him/her to be a paid employee, or (2) at which the researcher is a matriculated student. Scholars, faculty, fellows, and students who are visiting the UW and who are the lead researcher: identify your home institution and describe the purpose and duration of your UW visit, as well as the UW department/center with which you are affiliated while at the UW.

Note that many UW clinical faculty members are paid employees of non-UW institutions.

The UW IRB provides IRB review and oversight for only those researchers who meet the criteria described in the **SOP Use of the UW IRB**.

University of Washington

(1.2) Consultation history. Has there been any consultation with someone at HSD about this study?

It is not necessary to obtain advance consultation. However, if advance consultation was obtained, answering this question will help ensure that the IRB is aware of and considers the advice and guidance provided in that consultation.



→ If yes, briefly describe the consultation: approximate date, with whom, and method (e.g., by email, phone call, in-person meeting).

Elizabeth Falsberg and Jenny Maki IRB Reliance Administrator

: Discussion around reliance and that this is a just-in-time, funder requested application

**1.3** Similar and/or related studies. Are there any related IRB applications that provide context for the proposed activities?

Examples of studies for which there is likely to be a related IRB application: Using samples or data collected by another study; recruiting subjects from a registry established by a colleague's research activity; conducting Phase 2 of a multi-part project, or conducting a continuation of another study; serving as the data coordinating center for a multi-site study that includes a UW site.

Providing this information (if relevant) may significantly improve the efficiency and consistency of the IRB's review.



→ If yes, briefly describe the other studies or applications and how they relate to the proposed activities. If the other applications were reviewed by the UW IRB, please also provide: the UW IRB number, the study title, and the lead researcher's name.

**1.4** Externally-imposed urgency or time deadlines. Are there any externally-imposed deadlines or urgency that affect the proposed activity?

HSD recognizes that everyone would like their IRB applications to be reviewed as quickly as possible. To ensure fairness, it is HSD policy to review applications in the order in which they are received. However, HSD will assign a higher priority to research with externally-imposed urgency that is beyond the control of the researcher. Researchers are encouraged to communicate as soon as possible with their HSD staff contact person when there is an urgent situation (in other words, before submitting the IRB application). Examples: a researcher plans to test an experimental vaccine that has just been developed for a newly emerging epidemic; a researcher has an unexpected opportunity to collect data from students when the end of the school year is only four weeks away.

HSD may ask for documentation of the externally-imposed urgency. A higher priority should not be requested to compensate for a researcher's failure to prepare an IRB application in a timely manner. Note that IRB review requires a certain minimum amount of time; without sufficient time, the IRB may not be able to review and approve an application by a deadline.



 $\rightarrow$  If yes, briefly describe the urgency or deadline as well as the reason for it.

NIH is ready to issue Notice of Award pending IRB determination. Our NIH project officer has requested we include our IRB determination with our just in time materials.

**1.5 Objectives** Using lay language, describe the purpose, specific aims, or objectives that will be met by this specific project. If hypotheses are being tested, describe them. You will be asked to describe the specific procedures in a later section.

If this application involves the use of a HUD "humanitarian" device: describe whether the use is for "on-label" clinical patient care, "off-label" clinical patient care, and/or research (collecting safety and/or effectiveness data).

To test the preliminary efficacy of the Journey of Transformation—Native Youth Health Leadership Program (CHJ) which is an adapted and expanded version of the Discovering Our Story intervention curriculum, a 2010 SAMSHA-identified best practice AIAN strengths-based comprehensive substance use and health risk prevention and health leadership program for AIAN youth.

### Outcomes:

- decrease rates of ATOD (marijuana and other drugs) use, intentions to use, susceptibility,
- increase refusal efficacy;
- decrease sexual activity (number of partners, condomless intercourse
- delay sexual initiation,
- increase sexual self-efficacy (i.e., refusal, avoidance), and safer sex intentions.

Examine how stressful life events, mental health (depression/anxiety/self-esteem), cultural protective (identity, enculturation, collectivist values, community connectedness, communal mastery, benevolence/traditionalism) and PYD-related factors (e.g., connectedness, efficacy, ATOD and sexual refusal) moderate or mediate the intervention's efficacy.

(1.6) Study design. Provide a one-sentence description of the general study design and/or type of methodology.

Your answer will help HSD in assigning applications to reviewers and in managing workload. Examples: a longitudinal observational study; a double-blind, placebo-controlled randomized study; ethnographic interviews; web scraping from a convenience sample of blogs; medical record review; coordinating center for a multi-site study.

A randomized waitlist stepped wedge design with study participants recruited in staggered cohorts, with those in each annual recruitment wave receiving *individual-level random assignment* to either immediate intervention or waitlist control.

(1.7) Intent. Check all the descriptors that apply to your activity. You must place an "X" in at least one box.

This question is essential for ensuring that your application is correctly reviewed. Please read each option carefully.

| Descriptor |
|---|
| 1. Class project or other activity whose purpose is to provide an educational experience for the researcher (for example, to learn about the process or methods of doing research). |
| 2. Part of an institution, organization, or program's own internal operational monitoring. |
| 3. Improve the quality of service provided by a specific institution, organization, or program. |
| <ul> <li>4. Designed to expand the knowledge base of a scientific discipline or other scholarly field of study, and produce results that: <ul> <li>Are expected to be applicable to a larger population beyond the site of data collection or the specific subjects studied, or</li> <li>Are intended to be used to develop, test, or support theories, principles, and statements of relationships, or to inform policy beyond the study.</li> </ul> </li> </ul> |
| 5. Focus directly on the specific individuals about whom the information or biospecimens are collected through oral history, journalism, biography, or historical scholarship activities, to provide an accurate and evidence-based portrayal of the individuals. |
| 6. A quality improvement or program improvement activity conducted to improve the implementation (delivery or quality) of an accepted practice, or to collect data about the implementation of the practice for clinical, practical, or administrative purposes. This does not include the evaluation of the efficacy of different accepted practices, or a comparison of their efficacy. |
| 7. Public health surveillance activities conducted, requested, or authorized by a public health authority for the sole purpose of identifying or investigating potential public health signals or timely awareness and priority setting during a situation that threatens public health. |
| 8. Preliminary, exploratory, or research development activities (such as pilot and feasibility studies, or reliability/validation testing of a questionnaire) |
| 9. Expanded access use of a drug or device not yet approved for this purpose |
| 10. Use of a Humanitarian Use Device |

| 11. O | ther. Explain: |
|-------|----------------|

- **1.8** Background, experience, and preliminary work. Answer this question <u>only</u> if the proposed activity has one or more of the following characteristics. The purpose of this question is to provide the IRB with information that is relevant to its risk/benefit analysis.
  - Involves more than minimal risk (physical or non-physical)
  - Is a clinical trial, or
  - Involves having the subjects use a drug, biological, botanical, nutritional supplement, or medical device.

"Minimal risk" means that the probability and magnitude of harm or discomfort anticipated in the research are not greater than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests.

**a.** <u>Background</u>. Provide the rationale and the scientific or scholarly background for the proposed activity, based on existing literature (or clinical knowledge). Describe the gaps in current knowledge that the project is intended to address.

This should be a plain language description. Do not provide scholarly citations. Limit your answer to less than one page, or refer to an attached document with background information that is no more than three pages long.

Study is a phase 2 clinical trial.

Evidence shows that Native Americans have high rates of substance use disorder (ATOD) over the lifetime and die at higher rates than non-Natives from ATOD-related diseases such as cirrhosis and suicide. They also have a higher prevalence of behavioral risk factors for substance misuse and sexual health risk. AIAN youth are at the heart of this health crisis. AIAN youth have a lower overall mean age of tobacco use, alcohol use, and marijuana initiation (11.5 years) than the general population. Early initiation of ATOD use is associated with an array of negative physical and behavioral health outcomes including academic challenges, later ATOD abuse, and early sexual initiation. AIAN youth also have the earliest age of first sexual intercourse, and have more sexual partners than their non-AIAN counterparts. To stem the epidemic of ATOD-SRH-related health disparities among AIAN youth, collaborative partnerships must focus on development of culturally grounded, sustainable health interventions that incorporate healing related to historical trauma. In response, we will adapt and expand a promising Native-specific intervention, Discovering Our Story, to develop the Journey of Transformation (CJT) - Native Health Youth Leadership Program, an intervention to prevent ATOD use and SRH in AIAN youth attending boarding school. If successful, this project would have high relevance for boarding and tribal day school students across the country.

This research will fill an immediate gap in the substance use and sexual health risk (ATOD-SHR) prevention literature and policy given the dire need for empirical research to document a culturally relevant and comprehensive ATOD-SHR health promotion model. Data on the feasibility, acceptability, and efficacy of a youth health leadership intervention among ATOD-SHR risk AIAN youth would be a significant contribution to the substance abuse and sexual and reproductive health fields for AIANs as well as other groups. The data obtained in this study will form the basis for future large-scale efficacy studies with multiple tribal groups. The proposed work will make several distinctive contributions, including: (1) being the first ATOD-SHR study conducted at an Indian boarding school; (2) being the first study that specifically theorizes the role of trauma on ATOD-SRH risk outcomes among AIAN youth; (4) using an Indigenist theoretical model

and empirical measures that capture specific culturally-based factors such as historical trauma and community connectedness; (5) focusing on ATOD- SHR prevention issues among AIAN youth, a group at high risk for ATOD- SRH health disparities; (4) incorporating some of the same measures (behavioral) used in Strong Heart Study, Circle of Life HIV prevention among AIAN youth; and (5) incorporating an interdisciplinary and intertribal team approach with American Indian community members, leaders, and elders. Additionally, the project is significant because it builds upon an established relationship with a Native organization and is geared toward continued development of the research infrastructure and health treatment capacity.

Given the health risks to this population and the scarcity of research focused on their needs, combined with the potential risks to participants and the anticipated benefits to public and AIAN health, the proposed research and its potential risks are considered reasonable by the investigative team.

**b.** Experience and preliminary work. Briefly describe experience or preliminary work or data (if any) that you, your team, or your collaborators/co-investigators have that supports the feasibility and/or safety of this study.

It is not necessary to summarize all discussion that has led to the development of the study protocol. The IRB is interested only in short summaries about experiences or preliminary work that suggest the study is feasible and that risks are reasonable relative to the benefits. Examples: Your team has already conducted a Phase 1 study of an experimental drug which supports the Phase 2 study being proposed in this application; your team has already done a small pilot study showing that the reading skills intervention described in this application is feasible in an after-school program with classroom aides; your team has experience with the type of surgery that is required to implant the study device; the study coordinator is experienced in working with subjects who have significant cognitive impairment.

| This research will be conducted by PI Dr. Evans-Campbell (enrolled Snohomish Tribe) and co-I Dr. |
|---|
| Karina Walters (enrolled Choctaw Nation) who co-direct the Indigenous Wellness Research Institute (IWRI). |
| They are highly experienced indigenous researchers who have conducted intervention research in Native |
| communities for the last 15-20 years respectively serving as PI or Co-PI on over 30 federally-funded studies |
| with tribal communities and/or Native organizations The least intervention team, lead By |
| nas extensive expertise in conducting school-based interventions with Native youth. and her |
| team have worked extensively with middle and high school students including several projects with |
| students. |

The study builds on preliminary research from Drs Evans-Campbell and Walters:

Preliminary Feasibility, Acceptability, and Efficacy of an AIAN-based MI Intervention. Drs. Evans-Campbell and Walters in partnership with the Tulalip Tribes completed a 12-month intervention that had a culturally tailored, 5-session MI-based CVD prevention component (həli?dx<sup>w</sup> Project; aka Healthy Hearts-U01HL087322-05). The project successfully culturally adapted MI for CVD prevention, trained AIANs to implement the intervention, and conducted a preliminary feasibility and efficacy trial. Initial results indicated that participants enthusiastically embraced the MI component. Findings indicate that participants that completed all MI sessions engaged in more moderate intensity exercise greater than 30 minutes, maintained at 12-month follow-up; and that greater MI attendance was significantly associated with enhanced CVD health.

<u>Yappalli study (NIDA RO1 DA037176)</u>. Yappalli is an experiential, outdoor-based 3-month (with a 10 day walk on the Trail of Tears) substance abuse-obesity prevention RCT targeting at-risk adult Choctaw women. However, findings from two separate qualitative studies- have been completed to date- (study 1) analysis drew on two sources of qualitative data from Choctaw tribal members: 14 semi-structured interviews and two focus groups (N=9) and study 2 analysis drew on 35 Yappalli participants who had completed the intervention. Qualitative data suggests that inclusion of a culturally-tailored IMB approach and culturally derived health promotion model helped our participants begin working toward individualized

Discovery our story (DOS) pilots and evaluation. Led by the DOS is recognized by SAMHSA CDC as a best practice intervention to develop an age-appropriate middle-school age DOS curriculum. As part of the study, focus group sessions were held over three years at partner locations seeking feedback from Portland's AIAN community. The DOS curriculum originally focused on four primary areas: addictions, diabetes prevention, domestic violence, and mental health prevention. Pilot results indicated that the intervention: connected participants to culture and knowledge; instigated memories of teachings of relatives; identified positive behavioral actions; and provided hope and practical strategies for healthful living. The efficacy of storytelling as a teaching method was one of the strongest findings.

This study will be monitored in compliance with a Data Safety and Monitoring board.

**1.9 Supplements**. Check all boxes that apply, to identify relevant Supplements that should be completed and uploaded to *Zipline*.

This section is here instead of at the end of the form to reduce the risk of duplicating information in this IRB Protocol form that you will need to provide in these Supplements.

| Check all<br>That Apply | Type of Research | Supplement Name |
|---|---|---|
| | <b>Department of Defense</b> The research involves Department of Defense funding, facilities, data, or personnel. | SUPPLEMENT Department of Defense |
| | <b>Department of Energy</b> The research involves Department of Energy funding, facilities, data, or personnel. | SUPPLEMENT Department of Energy |
| | <b>Drug, biologic, botanical, supplement</b> Procedures involve the use of <u>any</u> drug, biologic, botanical or supplement, even if the item is not the focus of the proposed research | SUPPLEMENT Drugs |
| | Emergency exception to informed consent Research that requires this special consent waiver for research involving more than minimal risk | SUPPLEMENT Exception<br>from Informed Consent<br>for Emergency Research<br>(EFIC) |
| | Genomic data sharing Genomic data are being collected and will be deposited in an external database (such as the NIH dbGaP database) for sharing with other researchers, and the UW is being asked to provide the required certification or to ensure that the consent forms can be certified | SUPPLEMENT Genomic Data Sharing |
| | Medical device Procedures involve the use of <u>any</u> medical device, even if the device is not the focus of the proposed research, except when the device is FDA-approved and is being used through a clinical facility in the manner for which it is approved | SUPPLEMENT Devices |
| х | Multi-site or collaborative study The UW IRB is being asked to review on behalf of one or more non-UW institutions in a multi-site or collaborative study. | SUPPLEMENT Multi-site<br>or Collaborative Research |
| | | SUPPLEMENT Non-UW<br>Individual Investigators |
| Document Date & Vers | ion | Researcher Date & Version |

| | Non-UW Individual Investigators The UW IRB is being asked to review on behalf of one or more non-UW individuals who are not affiliated with another organization for the purpose of the research. | |
|---|---|---|
| | Other REDCap Installation Attestation for Electronic Consent The research will use a non-UW installation of REDCap for conducting and/or documenting informed consent. | SUPPLEMENT Other<br>REDCap Installation |
| | None of the above | |
| measures<br>essential<br>procedur<br>(d) no par<br>clinical vis<br>Review the | Confirm by checking the box below that you will comply with these basic COVID infection and risk control measures, OR that you have an exception granted by the HSD Director: (a) the only in-person interactions are essential for the study; (b) study team members and participants will wear face coverings throughout all procedures; (c) all study staff and participants will be screened for COVID-19 just prior to each research visit; and (d) no participants over the age of 85 years will be enrolled if their in-person participation is not connected with a clinical visit. See this webpage for details, including what "screening" means. Review the HSD website for current guidelines about which in-person research activities are allowable. | |
| 2 PARTICIF | ANTS | |
| | <b>ts</b> . Describe the general characteristics of the subject populations or groups, incealth status, and any other relevant characteristics. | cluding age range, |
| | outh, all genders (ages 13-16) attending the Indian School | |
| a. Inclusio | and exclusion criteria.<br>In criteria. Describe the specific criteria that will be used to decide who will be i<br>mong interested or potential subjects. Define any technical terms in lay languag | |
| (a) be<br>and | e youth must be:<br>tween 13 years of age and 16 years of age;<br>rrently attend Indian School in the 9 <sup>th</sup> grade. | |
| | on criteria. Describe the specific criteria that will be used to decide who will be the from subjects who meet the inclusion criteria listed above. Define any technic | |
| none | | |
| | IRB approval is required in order to include prisoners in research, even when parget population. | risoners are not an |
| Is the rese | arch likely to have subjects who become prisoners while participating in the stu | dy? |
| For example,<br>during the st | a longitudinal study of youth with drug problems is likely to have subjects who will be pudy. | risoners at some point |
| X No | | |

| Yes | • | ct becomes a prisoner while participating in the study, will any study procedures lection related to the subject be continued while the subject is a prisoner? |
|---|---|---|
| | No | rection related to the subject be continued while the subject is a prisoner. |
| | | If yes, describe the procedures and/or data collection that will continue with prisoner subjects |
| | Г | |
| <b>2.4</b> Will the prop | osed research recrui | it or obtain data from individuals that are known to be prisoners? |
| | - | do not indicate prisoner status and prisoners are not a target population, select "No". See definition of "prisoner". |
| X No<br>Yes | → If yes, answer th | ne following questions (i – iv). |
| | i. Describe the t | ype of prisoners, and which prisons/jails: |
| | general living<br>earnings in pr | about prisoner research is whether the effect of participation on prisoners' conditions, medical care, quality of food, amenities, and/or opportunity for rison will be so great that it will make it difficult for prisoners to adequately research risks. How will the chances of this be reduced? |
| | will be fair to | It will be done to make sure that (a) recruitment and subject selection procedures all eligible prisoners and (b) prison authorities or other prisoners will not be able prevent or require particular prisoners from participating. |
| | Washington (a) not encou<br>parole decision | h will involve prisoners in federal facilities or in state/local facilities outside of State: check the box below to provide assurance that study team members will trage or facilitate the use of a prisoner's participation in the research to influence ons, and (b) clearly inform each prisoner in advance (for example, in a consent articipation in the research will have no effect on his or her parole. |
| | Confirme | ed |
| for any of the | • | oval is required for the use of the subject populations listed here. Check the boxes will be purposefully included. (In other words, being a part of the population is y.) |
| The WORKSHE | EETS describe the criter | ria for approval but do not need to be completed and should not be submitted. |
| | Population | Worksheet |
| Fetuse | s in utero | WORKSHEET Pregnant Women |

| Neonates of uncertain viability | WORKSHEET Neonates |
|---|---|
| Non-viable neonates | WORKSHEET Neonates |
| Pregnant women | WORKSHEET Pregnant Women |
| a. If you check any of the boxes above, use to consider. | e this space to provide any information that may be relevant for the IRB |
| | <b>populations.</b> Will Native American or non-U.S. indigenous populations e-focused organization, or similar community-based organization? |
| | or national legislation as having a set of specific rights based on their historical or historical distinctiveness from other populations that are often politically |
| Examples: a reservation school or health clinic, | ; recruiting during a tribal community gathering |
| UW IRB expects that tribal,<br>This may or may not involv | al-focused organization, or similar community-based organization. The /indigenous approval will be obtained before beginning the research. we approval from a tribal IRB. The study team and any are also responsible for identifying any tribal laws that may affect the |
| | operated by the Bureau of Indian Affairs. It is not tribally owned or ort is provided by the principal see attachments. |
| partnership with the aspects of the project protecurriculum are appropriate We will formalize <b>two major</b> 1) Cultural and Scientific A expertise in positive youth | or community advisory groups-<br>Advisory Council (CSAC) The CSAC will include Native researchers with leadership interventions and experts in prevention science. |
| | <b>(YAC)</b> . The <i>Youth Advisory Council</i> will consist of 8 youth drawn from the oalition and other youth leadership groups on campus. The CSAC will |

meet 4 times per year and the YAC will convene monthly during the school year.

**2.7 Third party subjects.** Will the research collect private identifiable information about *other individuals* from the study subjects? Common examples include: collecting medical history information or contact information about family members, friends, co-workers.

"Identifiable" means any direct or indirect identifier that, alone or in combination, would allow you or another member of the research team to <u>readily identify</u> the person. For example, suppose that the research is about immigration history. If subjects are asked questions about their grandparents but are not asked for names or other information that would allow easy identification of the grandparents, then private identifiable information is not being collected about the grandparents and the grandparents are not subjects.

| X No | |
|---|---|
| Yes | → If yes, these individuals are considered human subjects in the study. Describe them and what data will be collected about them. |

**2.8 Number of subjects.** Is it possible to predict or describe the maximum number of subjects (or subject units) needed to complete the study, for each subject group?

<u>Subject units</u> mean units within a group. For most research studies, a group will consist of individuals. However, the unit of interest in some research is not the individual. Examples:

- Dyads such as caregiver-and-Alzheimer's patient, or parent and child
- Families
- Other units, such as student-parent-teacher

<u>Subject group</u> means categories of subjects that are meaningful for the specific study. Some research has only one subject group – for example, all UW students taking Introductory Psychology. Some common ways in which subjects are grouped include:

- By intervention for example, an intervention group and a control group.
- By subject population or setting for example, urban versus rural families
- By age for example, children who are 6, 10, or 14 years old.

The IRB reviews the number of subjects in the context of risks and benefits. Unless otherwise specified, if the IRB determines that the research involves no more than minimal risk: there are no restrictions on the total number of subjects that may be enrolled. If the research involves more than minimal risk: The number of enrolled subjects must be limited to the number described in this application. If it is necessary later to increase the number of subjects, submit a Modification. Exceeding the IRB-approved number (over-enrollment) will be considered non-compliance.

No → If no, provide the rationale in the box below. Also, provide any other available information about the scope/size of the research. You do not need to complete the table.

Example: It may not be possible to predict the number of subjects who will complete an online survey

advertised through Craigslist, but you can state that the survey will be posted for two weeks and the number who respond is the number who will be in the study.

→ If yes, for each subject group, use the table below to provide the estimate of the maximum desired number of individuals (or other subject unit, such as families) who will complete the research.

Group name/description

Maximum desired number of individuals (or other subject unit, such as families) who will complete the research

| | Provide numbers for the site(s) reviewed by the UW IRB and for the study-wide total number; example: 20/100 |
|---|---|
| Students | 450 |

**2.9 COVID-19 Screening**. If there will be any in-person interactions with the subjects, describe how you will screen them for COVID-19 symptoms within the 24 hours before the interaction. Also, describe the COVID-19 screening procedures for the study staff who will interact with the subjects.

Acceptable procedures include some type of symptom check or attestation, or a SARS-CoV-2 test with quick access to results. Symptom attestation involves an individual reviewing a list of symptoms and declaring the presence or absence of those symptoms. HSD strongly encourages adapting this Washington State Department of Health Screening Tool <a href="https://www.doh.wa.gov/Portals/1/Documents/1600/coronavirus/Employervisitorscreeningguidance.pdf">https://www.doh.wa.gov/Portals/1/Documents/1600/coronavirus/Employervisitorscreeningguidance.pdf</a> or the UW EH&S Example Symptom Self-Attestation in this document:

<u>https://www.ehs.washington.edu/system/files/resources/guidance-symptom-monitoring-COVID-19.pdf</u>. If you will test for the virus, you must also describe here whether the testing lab is CLIA-certified and how the results will be reported to the subjects.

We do not expect to engage human subjects till **Fall 2022**. If COVID concerns are still relevant at the time, we will follow the current CDC guidelines.

### 3 NON-UW RESEARCH SETTING

Complete this section only if UW investigators and people named in the <u>SUPPLEMENT:</u>

<u>Non-UW Individual Investigators</u> will conduct research procedures outside of UW and Harborview

**3.1**) Reason for locations. Describe the reason(s) for choosing the locations.

This is especially important when the research will occur in locations or with populations that may be vulnerable to exploitation. One of the three ethical principles the IRB must consider is justice: ensuring that reasonable, non-exploitative, and well-considered procedures are administered fairly, with a fair distribution of costs and potential benefits.

While there is a paucity of research addressing the substance use and sexual health risk prevention needs of Native youth in general, there is even less information available on substance use and sexual health-related health disparities for the nearly 1 out of 10 Native youth attending the 183 Indian schools in the US. If successful, this project would have high relevance for Native school students across the country.

**3.2**Local context. Culturally appropriate procedures and an understanding of local context are an important part of protecting subjects. Describe any site-specific cultural issues, customs, beliefs, or values that may affect the research, how it is conducted, or how consent is obtained or documented.

Examples: It would be culturally inappropriate in some international settings for a woman to be directly contacted by a male researcher; instead, the researcher may need to ask a male family member for permission before the woman can be approached. It may be appropriate to obtain permission from community leaders prior to obtaining consent from individual members of a group. In some distinct cultural groups, signing forms may not be the norm.

This federal site maintains an international list of human research standards and requirements: <a href="http://www.hhs.gov/ohrp/international/index.html">http://www.hhs.gov/ohrp/international/index.html</a>

As described in 2.6

- **3.3** Location-specific laws. Describe any local laws that may affect the research (especially the research design and consent procedures). The most common examples are laws about:
  - Specimens for example, some countries will not allow biospecimens to be taken out of the country.
  - **Age of consent** laws about when an individual is considered old enough to be able to provide consent vary across states, and across countries.
  - **Legally authorized representative** laws about who can serve as a legally authorized representative (and who has priority when more than one person is available) vary across states and countries.
  - Use of healthcare records many states (including Washington State) have laws that are similar to the federal HIPAA law but that have additional requirements.

| State: |
|---|
| A minor 15 years of age or older may give consent, without the consent of a parent or guardian of the minor, to: |
| (a) Hospital care, medical or surgical diagnosis or treatment by a physician licensed by the Medical Board |
| or a naturopathic physician licensed under ORS chapter 685, and dental or surgical diagnosis or treatment by a |
| dentist licensed by the Board of Dentistry, except as provided by ORS 109.660 (Construction). |
| (b) Diagnosis or treatment by a physician assistant who is licensed under ORS 677.505 (Application of provisions |
| governing physician assistants to other health professions) to 677.525 (Fees) and who is acting pursuant to a |
| practice agreement as defined in ORS 677.495 (Definitions for ORS 677.495 to 677.535). |
| (c)Diagnosis and treatment by a nurse practitioner who is licensed by the State Board of Nursing under |
| ORS 678.375 (Nurse practitioners) and who is acting within the scope of practice for a nurse practitioner. |
| (d)Except when the minor is obtaining contact lenses for the first time, diagnosis and treatment by an |
| optometrist who is licensed by the Board of Optometry under ORS 683.010 (Definitions for ORS 683.010 |
| to 683.310) to 683.340 (Duty to report prohibited conduct) and who is acting within the scope of practice for an |
| optometrist. [1971 c.381 §1; 2005 c.471 §7; 2010 c.91 §1; 2014 c.45 §11; 2017 c.356 §4] |
| A minor 14 years of age or older may obtain, without parental knowledge or consent, outpatient diagnosis or |
| treatment of a mental or emotional disorder or a chemical dependency, excluding methadone maintenance, by a |
| physician or physician assistant licensed by the Medical Board, a psychologist licensed by the |
| Board of Psychology, a nurse practitioner registered by the State Board of Nursing, a clinical social worker |
| licensed by the State Board of Licensed Social Workers, a professional counselor or marriage and family therapist |
| licensed by the Board of Licensed Professional Counselors and Therapists, a naturopathic physician |
| licensed by the Board of Naturopathic Medicine or a community mental health program established and |

operated pursuant to ORS 430.620 (Establishment of community mental health and developmental disabilities programs by one or more counties) when approved to do so by the Health Authority pursuant to rule. (2) However, the person providing treatment shall have the parents of the minor involved before the end of treatment unless the parents refuse or unless there are clear clinical indications to the contrary, which shall be documented in the treatment record. The provisions of this subsection do not apply to: (a)A minor who has been sexually abused by a parent; or (b) An emancipated minor, whether emancipated under the provisions of ORS 109.510 (Age of majority) and 109.520 (Majority of married persons) or 419B.550 (Definitions for ORS 419B.550 to 419B.558) to 419B.558 (Entry of judgment of emancipation) or, for the purpose of this section only, emancipated by virtue of having lived apart from the parents or legal guardian while being self-sustaining for a period of 90 days prior to obtaining treatment as provided by this section. [1985 c.525 §1; 1989 c.721 §47; 1993 c.546 §137; 1997 c.249 §38; 2009 c.442 §30; 2009 c.595 §71; 2013 c.178 §1; 2014 c.45 §13; 2017 c.6 §1; 2017 c.356 §6] **3.4)**Location-specific administrative or ethical requirements. Describe local administrative or ethical requirements that affect the research. Example: A school district may require researchers to obtain permission from the head district office as well as school principals before approaching teachers or students; a factory in China may allow researchers to interview factory workers but not allow the workers to be paid for their participation. Research must have permission from the School Principal before conducting research activities

| 3.5 If th | e PI is | a student: Does the research involve traveling outside of the US? |
|---|---|---|
| X | No | |
| | Yes | → If yes, confirm by checking the box that (1) you will register with the UW Office of Global Affairs |
| | _ | before traveling; (2) you will notify your advisor when the registration is complete; and (3) you will request a UW Travel Waiver if the research involves travel to the list of countries requiring a UW |
| | | Travel Waiver. |
| | | Confirmed |

# **4 RECRUITING and SCREENING PARTICIPANTS**

**4.1** Recruiting and Screening. Describe how subjects will be identified, recruited, and screened. Include information about: how, when, where, and in what setting. Identify who (by position or role, not name) will approach and recruit subjects, and who will screen them for eligibility.

Note: Per UW Medicine policy, the UW Medicine eCare/MyChart system may not be used for research recruitment purposes.

| • | before the start of the academic year, a short description about the study will be sent to freshman s/guardians in the school's new student package. The statement reads as follows: |
|---|---|
| 1. | CURRICULUM TESTING/DATA COLLECTION Initial for Consent: |
| | I (we) hereby grant permission/authorization for the above student to voluntarily participate in a research project testing a new Native American health curriculum highlighting youth leadership that uses traditional ways of teaching such as storytelling, making of drums, and story-vest |

making. Participation may include classroom activities, field trips, and online surveys about their connectedness to Native communities, relationships, and drug/alcohol use. Data gathered will determine how well this curriculum promotes leadership skills, Native cultural arts, connection to the natural environment, and how it promotes healthy decision-making around health and relationships.

2. Study Website (developed by UW staff)

the Website will provide the following information:

- A statement that the study involves research, an explanation of the purposes of the research, the expected duration of participation, a description of the procedures to be followed, and if applicable identification of any experimental procedures.
- A description of any foreseeable risks or discomforts to the subject
- A description of any benefits directly for the student or Native Communities that may be expected from the research.
- Information that if a student decides not to participate they will be offered any of the available current elective class options
- A statement describing the extent to which confidentiality, as well as information regarding mandatory
- Explanation of whom to contact for answers to pertinent questions about the research and their rights, and whom to contact in the event of a research-related harm.
- A statement that taking part in the study is voluntary, refusal to participate will involve no penalty or loss of benefits that the student is entitled and that they may discontinue participation at any time with no penalty or loss of benefits
- Information on the collection of identifiable information, when identifiers will be removed, and that the de-identified data could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from the student or guardian.
- 3. The Website will also provide a brief description with links to the full survey and assent form, as well as an Information Sheet that summarizes the information in the assent form in a Frequently Asked Questions (FAQ) format.
- 4. PI and PD will host informational ZOOM meetings. The parent study permission package and the Website will announce dates of monthly ZOOM informational meeting hosted by the PI and the Director. The ZOOM meetings will provide an overview of the study and respond to questions from guardians and students. 5. PI and PD contact information will be prominently placed on the website and they will be available to respond to individual inquires as requested. 6. Flyer (created by UW staff and distributed by UW staff and staff). A one page
- flyer will provide a brief description about the study, study curriculum content, note that the study is part of a research project, and instruct youth where they can find out more information. Contact information for the study team will also be included. The study flyer will be posted in the student newsletter, school student blog, and school parent newsletter.
- 7. Class presentation by UW staff and staff. Class presentations will be conducted in the spring and summer before the Fall trimester. Presentations are conducted by the Presentation will present similar content as on the Website and guardian permission document.

### Screening

All freshmen (9<sup>th</sup> grade) students at are American Indian or Alaska Native and between the ages of age of 13 and 16. Thus, by school administration assignment into the 9<sup>th</sup> grade student meet the recruitment criteria.

#### 4.2 Recruitment materials.

a. What materials (if any) will be used to recruit and screen subjects?

Examples: talking points for phone or in-person conversations; video or audio presentations; websites; social media messages; written materials such as letters, flyers for posting, brochures, or printed advertisements; questionnaires filled out by potential subjects.

Flyer

Study Website content

Class presentation talking points

Zoom Meetings talking points

We request flexibility to make minor revisions to our recruitment materials without submitting modifications to the IRB. If the revisions go outside the range and scope of approved materials and topics, we will submit a modification

**b.** Upload descriptions of each type of material (or the materials themselves) to **Zipline**. If letters or emails will be sent to any subjects, these should include a statement about how the subject's name and contact information were obtained. No sensitive information about the person (such as a diagnosis of a medical condition) should be included in the letter.

HSD encourages researchers to consider uploading descriptions of most recruitment and screening materials instead of the materials themselves. The goal is to provide the researchers with the flexibility to change some information on the materials without submitting a Modification for IRB approval of the changes. Examples:

- Provide a list of talking points that will be used for phone or in-person conversations instead of a script.
- For the description of a flyer, include the information that it will provide the study phone number and the name of a study contact person (without providing the actual phone number or name). This means that a Modification would not be necessary if/when the study phone number or contact person changes. Also, instead of listing the inclusion/exclusion criteria, the description below might state that the flyer will list one or a few of the major inclusion/exclusion criteria.
- For the description of a video or a website, include a description of the possible visual elements and a list of the content (e.g., study phone number; study contact person; top three inclusion/exclusion criteria; payment of \$50; study name; UW researcher).
- **4.3 Relationship with participant population**. Do any members of the study team have an existing relationship with the study population(s)?

Examples: a study team member may have a dual role with the study population (for example, being their clinical care provider, teacher, laboratory directory or tribal leader in addition to recruiting them for his/her research).



| Yes | → If yes, describe the nature of the relationship. |
|-----|----------------------------------------------------|

**4.4 Payment to participants**. The IRB must evaluate subject payment for the possibility that it will unduly influence subjects to participate. Refer to <u>GUIDANCE Subject Payment</u> when designing subject payment plans. Provide the following information about your plans for paying research subjects in the text box below or note that the information can be found in the consent form.

- The total amount/value of the payment
- Schedule/timing of the payment [i.e., when will subjects receive the payment(s)]
- Purpose of the payment [e.g., reimbursement, compensation, incentive]
- Whether payment will be "pro-rated" so that participants who are unable to complete the research may still receive some part of the payment

The IRB expects the consent process or study information provided to the subjects to include all of the above-listed information about payment, including the number and amount of payments, and especially when subjects can expect to receive payment. One of the most frequent complaints received by HSD is from subjects who expected to receive cash or a check on the day that they completed a study and who were angry or disappointed when payment took 6-8 weeks to reach them.

Participants will be paid up to \$75 for their time and effort for completing the follow-up assessments. They will be paid in the form of an online gift card after completing each assessment: \$20 for the second assessment; \$25 for the third assessment; and \$30 for the final assessment.

Because this project has been discontinued for this year, we are paying enrolled participants for completing the baseline assessment. We've been asked by the school principal to pay students who have finished the first survey since they will not go through the intervention or have the opportunity to take future surveys, and therefore receive compensation. The amount would be a \$20 online gift card, which is what they would be paid for the first follow-up assessment.

**4.5** Non-monetary compensation. Describe any non-monetary compensation that will be provided. Example: extra credit for students; a toy for a child. If class credit will be offered to students, there must be an alternate way for the students to earn the extra credit without participating in the research.

All youth in the class will receive project t-shirts, culturally relevant study posters, pens, writing pads, and water bottles for participation.

(4.6) Will data or specimens be accessed or obtained for recruiting and screening procedures prior to enrollment?

Examples: names and contact information; the information gathered from records that were screened; results of screening questionnaires or screening blood tests; Protected Health Information (PHI) from screening medical records to identify possible subjects.



No Yes → If no, skip the rest of this section; go to question 5.1.

→ If yes, describe the data and/or specimens (including PHI) and whether it will be retained as part of the study data.

**4.7 Consent for recruiting and screening**. Will consent be obtained for any of the recruiting and screening procedures? (Section 8: Consent of Adults asks about consent for the main study procedures).

"Consent" includes: consent from individuals for their own participation; parental permission; assent from children; consent from a legally authorized representative for adult individuals who are unable to provide consent.

#### Examples:

- For a study in which names and contact information will be obtained from a registry: the registry should have consent from the registry participants to release their names and contact information to researchers.
- For a study in which possible subjects are identified by screening records: there will be no consent process.
- For a study in which individuals respond to an announcement and call into a study phone line: the study team person talking to the individual may obtain non-written consent to ask eligibility questions over the phone.

| X No | → If no, skip the rest of this section; go to question 5.1. |
|---|---|
| Yes | s → If yes, describe the consent process. |
| | a. <u>Documentation of consent</u> . Will a written or verifiable electronic signature from the subject on a consent form be used to document consent for the <u>recruiting and screening procedures</u> ? |
| | No → If no, describe the information that will be provided during the consent process and for which procedures. |
| | Yes No and and the account form to 7 in line |
| | → If yes, upload the consent form to <b>Zipline</b> . |

# **5 PROCEDURES**

**5.1 Study procedures**. Using lay language, provide a complete description of the study procedures, including the sequence, intervention or manipulation (if any), drug dosing information (if any), blood volumes and frequency of draws (if any), use of records, time required, and setting/location. If it is available: Upload a study flow sheet or table to **Zipline**.

For studies comparing standards of care: It is important to accurately identify the research procedures. See UW IRB POLICY
Risks of Harm from Standard Care and the draft guidance from the federal Office of Human Research Protections, "Guidance on Disclosing Reasonably Foreseeable Risks in Research Evaluating Standards of Care"; October 20, 2014.

Information about pediatric blood volume and frequency of draws that would qualify for expedited review can be found in this reference table on the Seattle Children's IRB website.

Research activities will be conducted by UW and staff and begin the first week of class: for the waitlist group – the group starting in spring, they will only take the baseline assessment in the Fall and begin the intervention steps as described below beginning in the spring. Thus they receive one more assessment than students in the immediate intervention group (fall). UW staff will be on hand to answer any questions at each assessment time point. Please note the follow-up assessment are about 10 minutes shorter as we will not be any lifetime behaviors questions

Week 1. Take a 30-40 minute online baseline assessment.

UW and staff will set up laptops or students will have their own laptop. Students will be emailed a link, they will sign onto their laptops and link into the survey. The student

| will enter their response directly into the questionnaire. Students will be given a Native designed t-shirt |
|---|
| and water bottle. |
| Weeks 1-3. Meet with a mentor who will help students set goals to improve their health goals around sexual |
| health and/or reduce or avoid alcohol, tobacco, or other substance use. They may meet with the mentor |
| one more time within this time period (for a total of two meetings). The masters-level mentors are |
| provided by the analysis and trained by a certified motivational interviewer trainer |
| hired by UW. |
| Week 1 – 8 (month 1-2). As part of their health class, attend 16 health sessions related to healthy behaviors and |
| developing behavioral skills for health promotion. Sessions will be led by |
| staff. The study session curriculum will emphasize youth as leaders, storytellers, and environmental |
| stewards and highlight the importance of connecting to their own tribal traditions. |
| Week 9- 16 (month 3-4). <b>Optional</b> additional activity. Participate in once a month activity (booster sessions). The activities will help build youth leadership skills and include drum making, and storytelling vest making |
| that incorporate their own cultural symbols, and up to two outdoor activity field trips. The field trips are to |
| a places of cultural significance near the school and involve a 30-45 minute hike. Activities are between 1-2 |
| hours and delivered by the state of the stat |
| Week 9 (Month 3) take the online post intervention assessment via a link sent to their email address by |
| the UW staff |
| Week 16 (month 4) <b>Optional</b> additional activity. Meet with their mentor for a booster MI session to revise their |
| vows for health and community leadership. |
| Week 9 -24 (month 3 - 6). Optional additional activity. Attend a digital storytelling training and up to three |
| monthly planning sessions to prepare for digital storytelling leadership premiere night. Training and planning |
| sessions are 1-2 hours long and held after school. Students will be asked to create a digital story about a health |
| promotion activity of their choice for their community. Some examples may be an increase in cultural activities |
| though participating in traditional games, an increase in promoting healthy lifestyle by planting a traditional |
| garden or a medicine garden base on their own tribal plants. These activities are delivered by the UW and |
| staff. |
| Week 24 (Month 6) take the online follow-up assessment via a link sent to their email address by the |
| UW staff |
| Week 25 (Month 6): Optional additional activity. Attend a leadership premiere night, present their digital |
| stories and/or share a story that they have learned about health promotion and celebrate their health |
| leadership journey. |
| Help prepare the leadership night traditional feast and giveaway that will honor their community culture |
| and values. |
| Month 12: Take the online follow-up assessment via a link sent to their email address by the UW staff |
| Recordings. Does the research involve creating audio or video recordings? |
| X No → If no, go to <u>question 5.3.</u> |
| Yes → If yes, verify that you have described what will be recorded in 5.1 and answer question <b>a</b> . |
| a. Before recording, will consent for being recorded be obtained from subjects and any other |
| individuals who may be recorded? |
| No → If no, email <a href="mailto:hsdinfo@uw.edu">hsdinfo@uw.edu</a> before submitting this application in Zipline. |
| In the email, include a brief description of the research and a note that |
| individuals will be recorded without their advance consent. |

| | that are performed solely for research purposes or clinical scans that are modified for research purposes (for<br>gadolinium-based contrast agent when it is not required for clinical reasons). |
|---|---|
| X No → | If no, go to <u>question <b>5.4</b></u> . |
| ☐ Yes → | If yes, answer questions <b>a</b> through <b>c</b> . |
| a. De | escribe the MRI scan(s). Specifically: |
| • | What is the purpose of the scan(s)? Examples: obtain research data; safety assessment |
| • | associated with a research procedure. Which subjects will receive an MRI scan? |
| • | |
| _ | the scans will occur. For example: all subjects will undergo two MRI scans, six months apart. |
| b. Mi | RI facility. At which facility(ies) will the MRI scans occur? Check all that apply. |
| b. MI | UWMC Radiology/Imaging Services (the UWMC clinical facility) DISC Diagnostic Imaging Sciences Center (UWMC research facility) CHN Center for Human Neuroscience MRI Center (Arts & Sciences research facility) BMIC Biomolecular Imaging Center (South Lake Union research facility) Harborview Radiology/Imaging Services (the Harborview clinical facility) SCCA Imaging Services Northwest Diagnostic Imaging |
| b. Mi | UWMC Radiology/Imaging Services (the UWMC clinical facility) DISC Diagnostic Imaging Sciences Center (UWMC research facility) CHN Center for Human Neuroscience MRI Center (Arts & Sciences research facility) BMIC Biomolecular Imaging Center (South Lake Union research facility) Harborview Radiology/Imaging Services (the Harborview clinical facility) SCCA Imaging Services |
| c. Pe | UWMC Radiology/Imaging Services (the UWMC clinical facility) DISC Diagnostic Imaging Sciences Center (UWMC research facility) CHN Center for Human Neuroscience MRI Center (Arts & Sciences research facility) BMIC Biomolecular Imaging Center (South Lake Union research facility) Harborview Radiology/Imaging Services (the Harborview clinical facility) SCCA Imaging Services Northwest Diagnostic Imaging |
| c. Pe | UWMC Radiology/Imaging Services (the UWMC clinical facility) DISC Diagnostic Imaging Sciences Center (UWMC research facility) CHN Center for Human Neuroscience MRI Center (Arts & Sciences research facility) BMIC Biomolecular Imaging Center (South Lake Union research facility) Harborview Radiology/Imaging Services (the Harborview clinical facility) SCCA Imaging Services Northwest Diagnostic Imaging Other: identify in the text box below: |

**(5.4) Data variables.** Describe the specific data that will be obtained (including a description of the most sensitive items). Alternatively, a list of the data variables may be uploaded to *Zipline*.

These examples are of the most sensitive and risky questions we may ask. None of the measures are intended to capture information on suicidality or some other condition that would need referral or notification to some other entity. Please note the follow-up assessment are about 10 minutes shorter as we will not be collecting any lifetime behaviors questions.

Alcohol, Tobacco and Other Drug Use.

Current alcohol use. Participants will be asked if they drank alcohol in the past 30 days

Problem drinking, GAINS Short Screener for youth

ATOD Age initiation. Age of first alcohol, tobacco, marijuana and other drug use.

<u>Peer Alcohol Associations</u>. Number of friends that drink often, peer encouragement to drink or get drunk.<sup>42</sup> <u>Susceptibility to initiate ATOD</u> among self-reported non-smokers, non-drinkers, and non-drug users we will ask 6 questions on a 4-point scale: (eg. "If one of your best friends offered you a cigarette/joint/drink, would you smoke it?").

<u>Specific Event Drug and Alcohol Refusal Efficacy scale (SEDARE)</u> perceived likelihood that youth will use drugs and alcohol in specific situations and inquires whether the respondent would be tempted to use alcohol or marijuana in eight potentially stressful or pressured situations. <sup>43</sup>

<u>Non-ceremonial tobacco use</u>. Adapted from the NSDUH include current cigarette use, vaping and juuling. **Adolescent Sexual and Reproductive Health.** 

<u>Sexual activity</u>. Adolescent Sexual Risk Behavior 11-item and Adolescent Sexual Activity Index (ASAI) 10 items assess current and past sexual practices with most items focused on pre-coital behaviors during last 12 months for the sexual activities with other youth. If yes to pre-coital behaviors additional items assess if they have engaged in sexual intercourse, frequency, frequency of sex without birth control, frequency of sex without a condom; number of different sexual partners; and whether or not alcohol or drugs were used at first sex experience and/or last time had sex.

<u>Safer sex intentions</u>. Health Belief Model-Intentions for Safer Sex (HBMI) 7-item/5 pt scale (e.g., "I do not plan on having sex until I am at least 18 years old").

**Predictors, Mediators, and Moderators**. Spirituality (*Native American Spirituality Scale, Traditional Spiritual* Activities scale)

#### Standard measures:

Mental health/well-being (e.g., self-esteem, GAD-7, and PHQ-8) for youth and culturally-specific stressors such as familial historical trauma, microagressions, in-community microaggressions.

<u>Community Values Scale</u>, level of internalization of AIAN collective values related to traditionalism and benevolence.

Hemingway Measure of Adolescent Connectedness. 45 Positive Youth Development-related moderators.

**5.5 Data sources.** For all types of data that will be accessed or collected for this research: Identify whether the data are being obtained from the subjects (or subjects' specimens) or whether they are being obtained from some other source (and identify the source).

If you have already provided this information in Question 5.1, you do not need to repeat the information here.

All data collected will be from youth participants via the online survey

**5.6 Identifiability of data and specimens**. Answer these questions carefully and completely. This will allow HSD to accurately determine the type of review that is required and the relevant compliance requirements. Review the following definitions before answering the questions:

Access means to view or perceive data, but not to possess or record it. See, in contrast, the definition of "obtain". Identifiable means that the identity of an individual is or may be readily (1) ascertained by the researcher or any other member of the study team from specific data variables or from a combination of data variables, or (2) associated with the information.

**Direct identifiers** are direct links between a subject and data/specimens. Examples include (but are not limited to): name, date of birth, medical record number, email or IP address, pathology or surgery accession number, student number, or a collection of data that is (when taken together) identifiable.

**Indirect identifiers** are information that links between direct identifiers and data/specimens. Examples: a subject code or pseudonym.

**Key** refers to a single place where direct identifiers and indirect identifiers are linked together so that, for example, coded data can be identified as relating to a specific person. Example: a master list that contains the data code and the identifiers linked to the codes.

**Obtain** means to possess or record in any fashion (writing, electronic document, video, email, voice recording, etc.) for research purposes and to retain for any length of time. This is different from **accessing**, which means to view or perceive data.

| . will you or al | ny members of your team nave <u>access</u> to any direct or indirect identifiers? |
|---|---|
| X Yes | → If yes, describe which identifiers and for which data/specimens. |
| | will have access to students' names, email address, and phone numbers so they can engage students in the intervention. UW staff will have access to names, email address, and phone numbers and the link file so they can conduct longitudinal data collection. |
| No | → If no, select the reason(s) why you (and all members of your team) will not have access to direct or indirect identifiers. |
| | There will be no identifiers. |
| | Identifiers or the key have been (or will have been) destroyed before access. |
| | There is an agreement with the holder of the identifiers (or key) that prohibits the release of the identifiers (or key) to study team members under any circumstances. |
| | This agreement should be available upon request from the IRB. Examples: a Data Use Agreement, Repository Gatekeeping form, or documented email. |
| | There are written policies and procedures for the repository/database/data management center that prohibit the release of the identifiers (or identifying link). This includes situations involving an Honest Broker. |
| | There are other legal requirements prohibiting the release of the identifiers or key. Describe them below. |

| <b>b.</b> Will you or any st | tudy team members <u>obtain</u> any direct or indirect identifiers? |
|---|---|
| X Yes | ightarrow If yes, describe which identifiers and for which data/specimens. |
| | students' names, email address, and phone numbers so students can engage in the intervention. |
| No | → If no, select the reason(s) why you (and all members of your team) will not obtain direct or indirect identifiers. |
| | There will be no identifiers. |
| | Identifiers or the key have been (or will have been) destroyed before access. |
| | There will be an agreement with the holder of the identifiers (or key) that prohibits the release of the identifiers (or key) under any circumstances. |
| | This agreement should be available upon request from the IRB. Examples: a Data Use Agreement, Repository Gatekeeping form, or documented email. |
| | There are written policies and procedures for the repository/database/data management center that prohibit the release of the identifiers (or identifying link). This includes situations involving an Honest Broker. |
| | There are other legal requirements prohibiting the release of the identifiers or key. Describe them below. |
| • | will be obtained, indicate how the identifiers will be stored (and for which data). NOTE: Do data security plan here – that information is requested in section 9.6. |
| | Identifiers will be stored with the data. Describe the data to which this applies: |
| | Identifiers and study data will be stored separately but a link will be maintained between the identifiers and the study data (for example, through the use of a code). Describe the data to which this applies: |
| | Identifiers will be stored on a password protected Excel file on a password protected computer. |
| | Only UW research staff will facilitate data collection. The only connection between students' research data (assessments) and identifiers is a unique code stored on one file, on a secured server, password protected file. |
| | Identifiers and study data will be stored separately, with no link between the identifiers and the study data. Describe the data to which this applies: |

| | borator's institution/organization. |
|---|---|
| | ples include but are not limited to: (1) study, interpretation, or analysis of the data that results from the coded<br>nation or specimens; and (2) authorship on presentations or manuscripts related to this work. |
| no | |
| or any reas | <b>lealth Information (PHI).</b> Will participants' identifiable PHI be accessed, obtained, used, or disclose son (for example, to identify or screen potential subjects, to obtain study data or specimens, for sturbat does not involve the creation or obtaining of a Limited Data Set? |
| ntity" by fed<br><b>Jestion if t</b> l | ually identifiable healthcare record information or clinical specimens from an organization considered a "cover<br>deral HIPAA regulations, in any form or media, whether electronic, paper, or oral. <b>You must answer yes to thi</b><br>the research involves identifiable health care records (e.g., medical, dental, pharmacy, nursing, billing, etc.),<br>thealthcare information from a clinical department repository, or observations or recordings of clinical |
| X No | → If no, skip the rest of this question; go to question 5.8 |
| Yes | → If yes, answer all of the questions below. |
| | a. Describe the PHI and the reason for using it. Be specific. For example, will any "free text" field |
| | (such as physician notes) be accessed, obtained, or used? |
| | <b>b.</b> Is any of the PHI located in Washington State? |
| | No |
| | Yes |
| | c. Describe the pathway of how the PHI will be accessed or obtained, starting with the source/location and then describing the system/path/mechanism by which it will be identified accessed, and copied for the research. Be specific. For example: directly view records; search through a department's clinical database; submit a request to Leaf. |
| | d. For which PHI will subjects provide HIPAA authorization before the PHI is accessed, obtained and/or used? |
| | <u>Confirm by checking the box</u> that the UW Medicine <u>HIPAA Authorization</u> form maintained or |
| | Confirm by checking the box that the UW Medicine HIPAA Authorization form maintained or HSD website will be used to access, obtain, use, or disclose any UW Medicine PHI. Confirmed |

| | Provide the follo | owing assurances by checking the boxes. |
|---|---|---|
| | | m necessary amount of PHI to accomplish the purposes described in this will be accessed, obtained and/or used. |
| | law, for aut | not be reused or disclosed to any other person or entity, except as required by horized oversight of the research study, or for other research for which the use e of PHI would be permitted. |
| | | 'accounting for disclosures" requirement will be fulfilled, if applicable. See <a href="UW">UW</a> <a href="mailto:smpliance-policy #104">Dmpliance Policy #104</a> . |
| | | e reasonable safeguards to protect against identifying, directly or indirectly, any ny report of the research. |
| 5.8 Genomic data sh | naring. Will the re | esearch obtain or generate genomic data? |
| X No<br>Yes → | f yes, answer the | question below. |
| <u> </u> | a. Will genomic of database)? | data from this research be sent to a national database (for example, NIH's dbGaP |
| | No | |
| | Yes | → If yes, complete the <b>SUPPLEMENT Genomic Data Sharing</b> and upload it to <b>Zipline</b> . |
| 5.9 Whole genome s<br>sequencing? | sequencing. For r | research involving biospecimens: Will the research include whole genome |
| Whole genome sed exome sequence of | | cing of a human germline or somatic specimen with the intent to generate the genome or |
| X No<br>Yes | | |

- **5.10** Possible secondary use or sharing of information, specimens, or subject contact information. Is it likely that the obtained or collected information, specimens, or subject contact information will be used for any of the following:
  - Future research not described in this application (in other words, secondary research)
  - Submission to a repository, registry, or database managed by the study team, colleagues, or others for research purposes
  - Sharing with others for their own research

Please consider the broadest possible future plans and whether consent will be obtained now from the subjects for future sharing or research uses (which it may not be possible to describe in detail at this time). Answer YES even if future sharing or uses will use de-identified information or specimens. Answer NO if sharing is unlikely or if the only sharing will be through the NIH Genomic Data Sharing described in question 5.8.

Many federal grants and contracts now require data or specimen sharing as a condition of funding, and many journals require data sharing as a condition of publication. "Sharing" may include (for example): informal arrangements to share banked data/specimens with other investigators; establishing a repository that will formally share with other researchers through written agreements; or sending data/specimens to a third party repository/archive/entity such as the Social Science Open Access Repository (SSOAR), or the UCLA Ethnomusicology Archive.

| <br> |
|------|
| No |

**X** Yes  $\rightarrow$  If yes, answer all of the questions below.

**a.** Describe what will be stored for future use, including whether any direct or indirect (e.g., subject codes) identifiers will be stored.

De-identified assessment data will be stored.

**b.** Describe what will be shared with other researchers or with a repository/database/registry, including whether direct identifiers will be shared and (for specimens) what data will be released with the specimens.

De-identified assessment data.

**c.** Who will oversee and/or manage the sharing?

Indigenous Wellness Research Institute Director of Research and the PI

**d.** Describe the possible future uses, including limitations or restrictions (if any) on future uses or users. As stated above, consider the broadest possible uses.

Examples: data will be used only for cardiovascular research; data will not be used for research on population origins.

The study de-identified data will be available after publication of the main study manuscripts; other resources such as training manuals and curriculum will be available after demonstration of their efficacy. All requests from other researchers will be considered on a case-by-case basis by the study investigators and research partners. Researchers requesting access will have to submit a request in writing describing their qualifications including their certification by their local IRB, analytic plans and other uses of the data/resources, and plans to secure the confidentiality and safety of the data. They will be required to agree in writing that they will not share the data with others, will use it only for the research purpose(s) they delineated, and will return or destroy the data upon completion. In order to maintain protection of our participants' privacy, no directly identifying information will be shared with outside investigators. Given the sensitive nature of the data we are collecting including substance use and sexual

behavior among youth, we will not be creating a public access file.

If the UW study team or collaborators from this study use data for future analyses, a data set will be prepared in such a way that the data cannot be relinked to the direct identifiers and the study team could not identify any individuals from the combination of indirect identifiers (age, gender, etc.) in the data set.

For data shared according to NIH requirements, the data set will be prepared in such a way that any indirect identifiers shared are, in our opinion, unlikely to be able to be used to reidentify any individuals.

e. <u>Consent</u>. Will consent be obtained now from subjects for the secondary use, banking and/or future sharing?

X No Yes

→ If yes, be sure to include the information about this consent process in the consent form (if there is one) and in the answers to the consent questions in Section 8.

**f.** <u>Withdrawal</u>. Will subjects be able to withdraw their data/specimens from secondary use, banking or sharing?

No X Yes

→ If yes, describe how, and whether there are any limitations on withdrawal.

Example: data can be withdrawn from the repository but cannot be retrieved after they are released.

At any time before the end of the study, a participant may notify UW or study staff in writing that they would like their data removed from the secondary analysis file and we will honor that request.

g. <u>Agreements for sharing or release</u>. Confirm by checking the box that the sharing or release will comply with UW (and, if applicable, UW Medicine) policies that require a formal agreement with the recipient for release of data or specimens to individuals or entities other than federal databases.

Data Use Agreements or Gatekeeping forms are used for data; Material Transfer Agreements are used for specimens (or specimens plus data). Do not attach any template agreement forms; the IRB neither reviews nor approves them

X Confirmed

**5.11 Communication with subjects during the study**. Describe the types of communication (if any) the research team will have with already-enrolled subjects during the study. Provide a description instead of the actual materials themselves.

Examples: email, texts, phone, or letter reminders about appointments or about returning study materials such as a questionnaire; requests to confirm contact information.

Study staff will use email, texts, phone, and letters to remind participants about events, trainings, surveys/questionnaire as well as periodic requests to confirm contact information. We will also post information and updates on our study website and member only Facebook page.

**5.12 Future contact with subjects**. Is there a plan to retain any contact information for subjects so that they can be contacted in the future?



→ If yes, describe the purpose of the future contact, and whether use of the contact information will be limited to the study team; if not, describe who else could be provided with the contact information. Describe the criteria for approving requests for the information.

Examples: inform subjects about other studies; ask subjects for additional information or medical record access that is not currently part of the study proposed in this application; obtain another sample.

**5.13 Alternatives to participation.** Are there any alternative procedures or treatments <u>that might be advantageous</u> to the subjects?

If there are no alternative procedures or treatments, select "No". Examples of advantageous alternatives: earning extra class credit in some time-equivalent way other than research participation; obtaining supportive care or a standard clinical treatment from a health care provider instead of participating in research with an experimental drug.



→ If yes, describe the alternatives.

Any student not interested in the study will have the option to stay in the class, but will not be asked to complete surveys.

- **5.14 Upload to** *Zipline* all data collection forms (if any) that will be directly used by or with the subjects, and any scripts/talking points that will be used to collect the data. Do not include data collection forms that will be used to abstract data from other sources (such as medical or academic records), or video recordings.
  - **Examples**: survey, questionnaires, subject logs or diaries, focus group questions.
  - **NOTE:** Sometimes the IRB can approve the general content of surveys and other data collection instruments rather than the specific form itself. This prevents the need to submit a modification request for future minor changes that do not add new topics or increase the sensitivity of the questions. To request this general approval, use the text box below to identify the questionnaires/surveys/ etc. for which you are seeking this more general approval. Then briefly describe the scope of the topics that will be covered and the most personal and sensitive questions. The HSD staff person who screens this application will let you know whether this is sufficient or whether you will need to provide more information.
  - For materials that cannot be uploaded: upload screenshots or written descriptions that are sufficient to enable the IRB to understand the types of data that will be collected and the nature of the experience for the participant. You may also provide URLs (website addresses) or written descriptions below. Examples of materials that usually cannot be uploaded: mobile apps; computer-administered test; licensed and restricted standardized tests.
  - For data that will be gathered in an evolving way: This refers to data collection/questions that are not pre-determined but rather are shaped during interactions with participants in response to observations and responses made during those

interactions. If this applies to the proposed research, provide a description of the process by which the data collection/questions will be established during the interactions with subjects, how the data collection/questions will be documented, the topics likely to be addressed, the most sensitive type of information likely to be gathered, and the limitations (if any) on topics that will be raised or pursued.

### Use this text box (if desired) to provide:

- Short written descriptions of materials that cannot be uploaded, such as URLs
- A description of the process that will be used for data that will be gathered in an evolving way.
- The general content of questionnaires, surveys and similar instruments for which general approval is being sought. (See the **NOTE** bullet point in the instructions above.)

We will develop in REDCap an online survey data collection tool. Measures will consist of items noted in 5.4 above.

(5.15) SARS-CoV-2 testing. Will the subjects be tested for the SARS-CoV-2 coronavirus?

If the only testing is to screen the subjects (question 2.8), you do not need to answer this question



'es  $\rightarrow$  If yes:

- Name the testing lab
- Confirm that the lab and its use of this test is CLIA-certified or certified by the Washington State Department of Health
- Describe whether you will return the results to the participants and, if yes, who will do it and how (including any information you would provide to subjects with positive test results).

**5.16** Research equipment and COVID-19. Does you research involve any equipment that will be used on more than one subject that is not part of a clinical facility?

Examples: a computer tablet, a portable research ultra-sound device).



→ If yes: confirm by checking the box below that the disinfection and cleaning of the equipment will meet the enhanced UW Environmental Health & Safety requirements described here:

<a href="https://www.ehs.washington.edu/system/files/resources/cleaning-disinfection-protocols-covid-19.pdf">https://www.ehs.washington.edu/system/files/resources/cleaning-disinfection-protocols-covid-19.pdf</a>

Confirmed

# 6 CHILDREN (MINORS) and PARENTAL PERMISSION

**(6.1)Involvement of minors**. Does the research include minors (children)?

Minor or child means someone who has not yet attained the legal age for consent for the research procedures, as described in the applicable laws of the jurisdiction in which the research will be conducted. This may or may not be the same as the definition used by funding agencies such as the National Institutes of Health.

- In Washington State the generic age of consent is 18, meaning that anyone under the age of 18 is considered a child.
- There are some procedures for which the age of consent is much lower in Washington State.
- The generic age of consent may be different in other states, and in other countries

| | • | | generic age of consent may be unreferred mother states, and mother countries. |
|---|---|---|---|
| | No | $\rightarrow$ | If no, go to <u>Section 8</u> . |
| Х | Yes | $\rightarrow$ | If yes, provide the age range of the minor subjects for this study and the legal age for consent in the study population(s). If there is more than one answer, explain. |
| | | | Age 13-16: Legal age in is 18 All participants are treated as minors and we will obtain parental permission and student assent. |
| | Don' | t kn | This means is it not possible to know the age of the subjects. For example, this may be true for some research involving social media, the Internet, or a dataset that is obtained from another researcher or from a government agency. Go to <a href="Section 8">Section 8</a> . |
| | _ | | |

- 6.2 Parental permission. Parental permission means actively obtaining the permission of the parents. This is not the same as "passive" or "opt out" permission where it is assumed that parents are allowing their children to participate because they have been provided with information about the research and have not objected or returned a form indicating they don't want their children to participate.
  - **a.** Will parental permission be obtained for:

| X All of the research procedures | → Go to guestion 6.2b. |
|---|---|
| None of the research procedures | → Use the table below to provide justification, and skip question 6.2b. |
| Some of the research procedures | → Use the table below to identify the procedures for which parental permission will not be obtained. |

Be sure to consider all research procedures and plans, including screening, future contact, and sharing/banking of data and specimens for future work.

| Will parents be informed about the research? <sup>3</sup> |
|-----------------------------------------------------------|
| NO |

Document Date & Version 01/21/2021

| able footnotes If the answer is the same for all children groups or all procedures: collapse the answer across the groups and/or procedures. If identifiable information or biospecimens will be obtained without parent permission, any waiver granted by the IRB does no override parents' refusal to provide broad consent (for example, through the Northwest Biotrust). Will parents be informed about the research beforehand even though active permission is not being obtained? b. Indicate the plan for obtaining parental permission. One or both boxes must be checked. Both parents, unless one parent is deceased, unknown, incompetent, or not reasonably available; or when only one parent has legal responsibility for the care and custody of the child \times One parent, even if the other parent is alive, known, competent, reasonably available, and shares legal responsibility for the care and custody of the child. This is all that is required for minimal risk research. If both boxes are checked, explain: X No Yes Yes, an advocate may need to be appointed for each child who is a ward. The advocate must be in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: • Background and experience • Willingness to act in the best interests of the child for the duration of the research • Independence of the research, research team, and any guardian organization | | |
|---|---|---|
| able footnotes If the answer is the same for all children groups or all procedures: collapse the answer across the groups and/or procedures. If identifiable information or biospecimens will be obtained without parent permission, any waiver granted by the IRB does no override parents' refusal to provide broad consent (for example, through the Northwest Biotrust). Will parents be informed about the research beforehand even though active permission is not being obtained? b. Indicate the plan for obtaining parental permission. One or both boxes must be checked. ■ Both parents, unless one parent is deceased, unknown, incompetent, or not reasonably available; or when only one parent has legal responsibility for the care and custody of the child ▼ One parent, even if the other parent is alive, known, competent, reasonably available, and shares legal responsibility for the care and custody of the child. This is all that is required for minimal risk research. If both boxes are checked, explain: ■ No Yes → If yes, an advocate may need to be appointed for each child who is a ward. The advocate must be in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: ■ Background and experience ● Willingness to act in the best interests of the child for the duration of the research | | |
| able footnotes If the answer is the same for all children groups or all procedures: collapse the answer across the groups and/or procedures. If identifiable information or biospecimens will be obtained without parent permission, any waiver granted by the IRB does no override parents' refusal to provide broad consent (for example, through the Northwest Biotrust). Will parents be informed about the research beforehand even though active permission is not being obtained? b. Indicate the plan for obtaining parental permission. One or both boxes must be checked. ■ Both parents, unless one parent is deceased, unknown, incompetent, or not reasonably available; or when only one parent has legal responsibility for the care and custody of the child ▼ One parent, even if the other parent is alive, known, competent, reasonably available, and shares legal responsibility for the care and custody of the child. This is all that is required for minimal risk research. If both boxes are checked, explain: ■ No Yes → If yes, an advocate may need to be appointed for each child who is a ward. The advocate must be in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: ■ Background and experience ● Willingness to act in the best interests of the child for the duration of the research | | |
| b. Indicate the plan for obtaining parental permission. One or both boxes must be checked. Both parents, unless one parent is deceased, unknown, incompetent, or not reasonably available; or when only one parent has legal responsibility for the care and custody of the child One parent, even if the other parent is alive, known, competent, reasonably available, and shares legal responsibility for the care and custody of the child. This is all that is required for minimal risk research. If both boxes are checked, explain: X No Yes → If yes, an advocate may need to be appointed for each child who is a ward. The advocate must be in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: Background and experience Willingness to act in the best interests of the child for the duration of the research | If the answer | :<br>r is the same for all children groups or all procedures: collapse the answer across the groups and/or procedures.<br>e information or biospecimens will be obtained without parent permission, any waiver granted by the IRB does no |
| Both parents, unless one parent is deceased, unknown, incompetent, or not reasonably available; or when only one parent has legal responsibility for the care and custody of the child One parent, even if the other parent is alive, known, competent, reasonably available, and shares legal responsibility for the care and custody of the child. This is all that is required for minimal risk research. If both boxes are checked, explain: A Children who are wards. Will any of the children be wards of the State or any other agency, institution, or entity? A No Yes If yes, an advocate may need to be appointed for each child who is a ward. The advocate must be in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: Background and experience Willingness to act in the best interests of the child for the duration of the research | | |
| only one parent has legal responsibility for the care and custody of the child One parent, even if the other parent is alive, known, competent, reasonably available, and shares legal responsibility for the care and custody of the child. This is all that is required for minimal risk research. If both boxes are checked, explain: Solution who are wards. Will any of the children be wards of the State or any other agency, institution, or entity? No Yes If yes, an advocate may need to be appointed for each child who is a ward. The advocate must be in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: Background and experience Willingness to act in the best interests of the child for the duration of the research | <b>b.</b> Indicate t | the plan for obtaining parental permission. One or both boxes must be checked. |
| responsibility for the care and custody of the child. This is all that is required for minimal risk research. If both boxes are checked, explain: 3 Children who are wards. Will any of the children be wards of the State or any other agency, institution, or entity? X No Yes If yes, an advocate may need to be appointed for each child who is a ward. The advocate must be in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: Background and experience Willingness to act in the best interests of the child for the duration of the research | | |
| This is all that is required for minimal risk research. If both boxes are checked, explain: 3 Children who are wards. Will any of the children be wards of the State or any other agency, institution, or entity? X No Yes → If yes, an advocate may need to be appointed for each child who is a ward. The advocate must be in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: ■ Background and experience ■ Willingness to act in the best interests of the child for the duration of the research | 1 1 | onsibility for the care and custody of the child. |
| As Children who are wards. Will any of the children be wards of the State or any other agency, institution, or entity? X No Yes → If yes, an advocate may need to be appointed for each child who is a ward. The advocate must be in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: Background and experience Willingness to act in the best interests of the child for the duration of the research | This is | |
| Yes → If yes, an advocate may need to be appointed for each child who is a ward. The advocate must be in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: Background and experience Willingness to act in the best interests of the child for the duration of the research | If b | ooth boxes are checked, explain: |
| Yes → If yes, an advocate may need to be appointed for each child who is a ward. The advocate must be in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: • Background and experience • Willingness to act in the best interests of the child for the duration of the research | | |
| Yes → If yes, an advocate may need to be appointed for each child who is a ward. The advocate must be in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: Background and experience Willingness to act in the best interests of the child for the duration of the research | .3 Children wh | no are wards. Will any of the children be wards of the State or any other agency, institution, or entity? |
| <ul> <li>Background and experience</li> <li>Willingness to act in the best interests of the child for the duration of the research</li> </ul> | VINA | |
| | V | in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The |
| | V | in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following points: |
| | V | <ul> <li>in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards.</li> <li>Describe who will be the advocate(s). The description must address the following points: <ul> <li>Background and experience</li> <li>Willingness to act in the best interests of the child for the duration of the research</li> </ul> </li> </ul> |
| | V | <ul> <li>in addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards.</li> <li>Describe who will be the advocate(s). The description must address the following points: <ul> <li>Background and experience</li> <li>Willingness to act in the best interests of the child for the duration of the research</li> </ul> </li> </ul> |

**6.4 UW Office for Youth Programs Development and Support.** If the project involves interaction (in-person or remotely) with individuals under the age of 18, researchers must comply with **UW Administrative Policy Statement 10.13** and the requirements listed at <a href="this website">this website</a>. This includes activities that are deemed to be Not Research or Exempt. It does not apply to third-party led research (i.e., research conducted by a non-UW PI). <a href="Information and FAQs">Information and FAQs</a> for researchers are available.

This point is advisory only; there is no need to provide a response.

# 7 ASSENT OF CHILDREN (MINORS)

Go to Section 8 if your research does not involve children (minors).

- **7.1** Assent of children (minors). Though children do not have the legal capacity to "consent" to participate in research, they should be involved in the process if they are able to "assent" by having a study explained to them and/or by reading a simple form about the study, and then giving their verbal choice about whether they want to participate. They may also provide a written assent if they are older. See <a href="WORKSHEET Children">WORKSHEET Children</a> for circumstances in which a child's assent may be unnecessary or inappropriate.
  - a. Will assent be obtained for:

| X All research procedures and child groups | → Go to question 7.2. |
|---|---|
| None of the research procedures and child groups | → Use the table below to provide justification, then skip to question <b>7.6</b> |
| Some of your research procedures and child groups | Use the table below to identify the procedures for which assent will not be obtained. |

Be sure to consider all research procedures and plans, including screening, future contact, and sharing/banking of data and specimens for future work.

| Children Group <sup>1</sup> | data/specimen collection (if any) for which assent will NOT be obtained | Reason why assent will not be obtained |
|---|---|---|
| <br> | | |

### Table footnotes

- 1. If the answer is the same for all children groups or all procedures, collapse your answer across the groups and/or procedures.
- **7.2 Assent process.** Describe how assent will be obtained, for each child group. If the research involves children of different ages, answer separately for each group. If the children are non-English speakers, include a description of how their comprehension of the information will be evaluated.

For students whose parent/guardian indicated they have permission to take the class, they will be invited to attend a research orientation meeting during their onsite school orientation. Students arrive to the school two weeks before classes start to move into their dorms, settle in, learn about class topics for the year and school activities. A research orientation session will occur during the first week of their 2-week pre-school orientation period.

At the orientation meeting, a study package will be handed to each youth. The package will include Native items such as sage or lavender, a writing pad and pen and pencil with a Native design and study phone number, two copies of the assent form (one for them to sign and the other to keep as their copy), and the study flyer. UW and staff will inform the students about the research project, highlighting that it is

| | completely voluntary and then review the assent form and ask for questions. At the end of the meeting, students will be instructed to write their names on the assent form and indicate if they are interested in participating in the project (Yes/No) or would like more information. Students who are interested in participating will also be asked to fill out a contact information sheet, which asks for their name(s), birth date, preferred pronouns, email address, phone number, and space to provide any additional contact information (ex., social media). If they would like more information, they will be asked to provide contact information (similar to that of those who have assented) and a UW staff person will contact them. They will be informed that they may also reach out to the UW or staff person will contact them before the first day of class (within the two weeks) if they have any additional questions about participation. |
|---|---|
| | Students will hand in one signed copy of the assent form when they exit the room. |
| | UW or staff will then follow-up with students that indicated they are interested in participating and welcome them to the program and asked if they have any additional questions. They will also follow-up with students who request additional information. |
| | For students that have indicated they are interested, they will be randomly assigned to a class offering the intervention sessions. Some classes will start the intervention curriculum in the Fall, others in the Spring. Students that indicated they are not interested they will be assigned to a class that is not participating in the intervention curriculum. This is easily done as there are multiple classes for each grade. |
| | Students may choose to drop out of the research program by notifying research staff by email and reassignment to a health class will be provided. As standard practice, students periodically change class assignments so this would not seem out of the norm. |
| | <b>Dissent or resistance.</b> Describe how a child's objection or resistance to participation (including non-verbal indications) will be identified during the research, and what the response will be. |
| | Turn in an assent form without a name or marked "no, not interested." |
| | Over the course of the 6-month program, participants may decline further participation by sending an email to the study team email address. All communication and all documents will provide a reminder that participation is voluntary. |
| | <b>7.4 E-consent.</b> Will any electronic processes (email, websites, electronic signatures, etc.) be used to present assent information to subjects/and or to obtain documentation (signatures) of assent? If yes, describe how this will be done. |
| | information to subjects/and or to obtain documentation (signatures) of assent? If yes, describe how this will be |
| | information to subjects/and or to obtain documentation (signatures) of assent? If yes, describe how this will be |
| 7.5 ( | information to subjects/and or to obtain documentation (signatures) of assent? If yes, describe how this will be done. |
| 7.5 ( | information to subjects/and or to obtain documentation (signatures) of assent? If yes, describe how this will be done. no Documentation of assent. Which of the following statements describes whether documentation of assent will be |
| 7.5 ( | information to subjects/and or to obtain documentation (signatures) of assent? If yes, describe how this will be done. no Documentation of assent. Which of the following statements describes whether documentation of assent will be obtained? None of the research procedures and child groups. Use the table below to provide justification, |

| | question <b>7.5.a</b> |
|---|---|
| <br>Children<br>Group¹ | Describe the procedures or data/specimen collection (if any) for which assent will NOT be documented |
| <br> | |
| <br> | |
| <br> | |

→ Complete the table below and then to go

### Table footnotes

- 1. If the answer is the same for all children groups or all procedures, collapse the answer across the groups and/or procedures.
  - **a. Describe how assent will be documented**. If the children are functionally illiterate or are not fluent in English, include a description of the documentation process for them.

All students attending the school in the 9<sup>th</sup> grade are literate and fluent in English. Documentation is their signature on the assent form.

- **b.** Upload all assent materials (talking points, videos, forms, etc.) to **Zipline**. Assent materials are not required to provide all of the standard elements of adult consent; the information should be appropriate to the age, population, and research procedures. The documents should be in Word, if possible.
- 7.6 Children who reach the legal age of consent during participation in longitudinal research.

<u>Children who were enrolled at a young age and continue for many years</u>: It is best practice to re-obtain assent (or to obtain it for the first time, if it was not obtained at the beginning of their participation).

<u>Children who reach the legal age of consent</u>: Informed consent must be obtained from the now-adult subject for (1) any ongoing interactions or interventions with the subjects, or (2) the continued analysis of specimens or data for which the subject's identify is readily identifiable to the researcher, unless the IRB waives this requirement.

a. Describe the plans (if any) to re-obtain assent from children.

The week before the Spring semester, students in the second wave will be emailed a welcome reminder about their upcoming spring research class. The reminder will include the study email address, study phone number, a copy of an assent form, a reminder their participation is voluntary, and a reminder that if they have any questions to please contact staff at the contact information provided (study email and phone is monitored by the UW staff). On the first day of Spring class, UW and staff will go to the study classes to review the assent forms, the study email address, study phone number, highlight that participation is voluntary, and ask students if they have any questions to please contact staff with the contact information provided.

- **b.** Describe the plans (if any) to obtain consent for children who reach the legal age of consent.
  - If adult consent will be obtained from them, describe what will happen regarding now-adult subjects who cannot be contacted.
  - If consent will not obtained or will not be possible: explain why.

Age range of children are 13-16. It will be impractical to obtain consent for continued data analysis when the minor participants turn 18.

- **7.7 Other regulatory requirements**. (This is for information only; no answer or response is required.) Researchers are responsible for determining whether their research conducted in schools, with student records, or over the Internet comply with permission, consent, and inspection requirements of the following federal regulations:
  - PPRA Protection of Pupil Rights Amendment
  - FERPA Family Education Rights and Privacy Act
  - COPPA Children's Online Privacy Protection Act

| CON |
|-----|

| Review the following definitions before answering the questions in this section. | | | |
|---|---|--|--|
| CONSENT | is the <u>process</u> of informing potential subjects about the research and asking them whether they want to participate. It does not necessarily include the signing of a consent form. | | |
| CONSENT<br>DOCUMENTATION | refers to how a subject's decision to participate in the research is documented. This is typically obtained by having the subject sign a consent form. | | |
| CONSENT FORM | is a document signed by subjects, by which they agree to participate in the research as described in the consent form and in the consent process. | | |
| ELEMENTS OF CONSENT | are specific information that is required to be provided to subjects. | | |
| CHARACTERISTICS OF<br>CONSENT | <ul> <li>are the qualities of the consent process as a whole. These are:</li> <li>Consent must be legally effective.</li> <li>The process minimizes the possibility of coercion or undue influence.</li> <li>Subjects or their representatives must be given sufficient opportunity to discuss and consider participation.</li> <li>The information provided must: <ul> <li>Begin with presentation of key information (for consent materials over 2,000 words)</li> <li>Be what a reasonable person would want to have</li> <li>Be organized and presented so as to facilitate understanding</li> <li>Be provided in sufficient detail</li> <li>Not ask or appear to ask subjects to waive their rights</li> </ul> </li> </ul> | | |
| PARENTAL PERMISSION | is the parent's active permission for the child to participate in the research. Parental permission is subject to the same requirements as consent, including written documentation of permission and required elements. | | |
| SHORT FORM CONSENT | is an alternative way of obtaining written documentation of consent that is most commonly used with individuals who are illiterate or whose language is one for which translated consent forms are not available. | | |
| | means there is IRB approval elements of consent in the c | for not obtaining consent or for not inclu<br>onsent process. | ding some of the | |
|---|---|---|---|--|
| WAIVER OF CONSENT NOTE: If you plan to obtain identifiable information or identifiable biospec consent, any waiver granted by the IRB does not override a subject's refus broad consent (for example, the Northwest Biotrust). | | | | |
| WAIVER OF | | | | |
| DOCUMENTATION OF CONSENT | • | oval for not obtaining written documenta | ation of consent. | |
| <b>8.1 Groups</b> Identify the gro | oups to which the answers in th | is section apply. | | |
| Adult subjects X Parents who are | providing permission for their | children to participate in research | | |
| | | " below should also be interpreted as app<br>erpreted as applying to the parents. | olying to parental | |
| | nd characteristics. This series outing and screening and, if yes | f questions is about whether consent will<br>, how. | be obtained for all | |
| to question 4.6. | | addressed in <u>question 4.7</u> . You do not need t | o repeat your answer | |
| <b>a</b> . Are there any proce | edures for which consent will no | ot be obtained? | | |
| | use the table below to identify to come studentify to the come student answer for some students. | the procedures for which consent will no<br>lies. | t be obtained. "All" | |
| Be sure to consider all res future work. | earch procedures and plans, includ | ding future contact, and sharing/banking of d | ata and specimens for | |
| Group <sup>1</sup> data/sp | ribe the procedures or<br>ecimen collection (if any)<br>n there will be NO consent<br>process | Reason why consent will not be obtained | Will subjects be provided with info about the research after they finish? | |

#### Table footnotes

- 1. If the answer is the same for all groups, collapse your answer across the groups and/or procedures.
  - **b.** <u>Describe the consent process</u>, if consent will be obtained for any or all procedures, for any or all groups. Address groups and procedures separately if the consent processes are different.

Be sure to include:

- The location/setting where consent will be obtained
- Who will obtain consent (refer to positions, roles, or titles, not names)
- How subjects will be provided sufficient opportunity to discuss the study with the research team and consider participation

#### **Parent Permission**

- 1. Parental Permission: We are asking for a waiver of documentation of parental permission. As per standard school policy the spring before Fall trimester begins, all parents are mailed a new student packet with an overview of the study. The overview includes a check box for parents/ guardians to indicate if they give their permission to invite their child to the project, study contact information, website and links for addition information. The study documents are written at the same language level as other information shares with parents.
- 2. The <u>parent permission information form</u> will be located on the website, access via the link, and sent via mail. It is attached.

For parents/guardians or students who may want more clarification, or have questions they also may:

- -Attend an informational ZOOM/video conferencing meeting offered by study staff. The guardian permission package and the Website will announce dates of monthly ZOOM informational meeting hosted by the PI and the Director. The ZOOM meetings will provide an overview of the study and respond to questions from guardians and students. The Zoom meeting platform is a standard form of communication between administrators, teachers, and parents.
- -Contact the PI and PD directly via the contact information prominently placed on the permission form and website. The PI and PD will be available to respond to individual inquiries as requested. All forms of communication will include a statement that taking part in the study is voluntary, refusal to participate will involve no penalty or loss of benefits that the student is entitled to, and that they may discontinue participation at any time with no penalty or loss of benefits.
- **c.** <u>Comprehension</u>. Describe the methods that will be used to ensure or test the subjects' understanding of the information during the consent process.
  - -All information will be written at the language level the school uses on their other documents and permission forms
  - -We will host informational ZOOM/video conferencing meetings.
  - The PI and site PI contact information (phone and email) will be prominently placed on the permission form and website and available to respond to individual inquiries as requested.

**d.** <u>Influence</u>. Does the research involve any subject groups that might find it difficult to say "no" to participation because of the setting or their relationship with someone on the study team, even if they aren't pressured to participate?

Examples: Student participants being recruited into their teacher's research; patients being recruited into their healthcare provider's research, study team members who are participants; outpatients recruited from an outpatient surgery waiting room just prior to their surgery.



→ If yes, describe what will be done to reduce any effect of the setting or relationship on the participation decision.

Examples: a study coordinator will obtain consent instead of the subjects' physician; the researcher will not know which subjects agreed to participate; subjects will have two days to decide after hearing about the study.

e. <u>Information provided is tailored to needs of subject population</u>. Describe the basis for concluding that the information that will be provided to subjects (via written or oral methods) is what a *reasonable member of the subject population(s)* would want to know. If the research consent materials contain a key information section, also describe the basis for concluding that the information presented in that section is that which is *most likely* to assist the selected subject population with making a decision. See <u>GUIDANCE Key Information for Consent Materials</u>.

For example: Consultation with publications about research subjects' preferences, disease-focused nonprofit groups, patient interest groups, or other researchers/study staff with experience with the specific population. It may also involve directly consulting selected members of the study population.

Permission form will be in the same format and language level as the school has always used thus both familiar and acceptable to the guardian population. We add in the option of video conference meetings-- a familiar form of school communication with guardians. We also provide and research staff contact information for one-to-one communication as desired/requested.

**f.** Ongoing process. For research that involves multiple or continued interaction with subjects over time, describe the opportunities (if any) that will be given to subjects to ask questions or to change their minds about participating.

Over the course of the 6-month program, participants may decline further participation, all communication documents provide a reminder that participation is voluntary. Parents may email or call the PI or PD via the contact information listed on the permission form and the website.

**8.3 Electronic presentation of consent information.** Will any part of the consent-related information be provided electronically for some or all of the subjects?

This refers to the use of electronic systems and processes instead of (or in addition to) a paper consent form. For example, an emailed consent form, a passive or an interactive website, graphics, audio, video podcasts. See <u>GUIDANCE Electronic Informed Consent</u> for information about electronic consent requirements at UW.

APPLICATION IRB Protocol



No

→ If no, skip to question 8.4

| If yes, answer questions <b>a</b> through <b>e</b> |
|---|
| <b>a</b> . Describe the electronic consent methodology and the information that will be provided. |
| All informational materials must be made available to the IRB. Website content should be provided as a Word document. It is considered best practice to give subjects information about multi-page/multi-screen information that will help them assess how long it will take them to complete the process. For example, telling them that it will take about 15 minutes, or that it involves reading six screens or pages. |
| <b>b.</b> Describe how the information can be navigated (if relevant). For example, will the subject be able to proceed forward or backward within the system, or to stop and continue at a later time? |
| c. In a standard paper-based consent process, the subjects generally have the opportunity to go<br>through the consent form with study staff and/or to ask study staff about any question they may<br>have after reading the consent form. Describe what will be done, if anything, to facilitate the<br>subject's comprehension and opportunity to ask questions when consent information is<br>presented electronically. Include a description of any provisions to help ensure privacy and<br>confidentiality during this process. |
| Examples: hyperlinks, help text, telephone calls, text messages or other type of electronic messaging, video conference, live chat with remotely located study team members. |
| d. What will happen if there are individuals who wish to participate but who do not have access to<br>the consent methodology being used, or who do not wish to use it? Are there alternative ways in<br>which they can obtain the information, or will there be some assistance available? If this is a<br>clinical trial, these individuals cannot be excluded from the research unless there is a compelling<br>rationale. |
| For example, consider individuals who lack familiarity with electronic systems, have poor eyesight or impaired motor skills, or who do not have easy email or internet access. |
| e. How will the research team ensure continued accessibility of consent materials and information<br>during the study? |
| f. How will additional information be provided to subjects during the research, including any |

| that allows v | Documentation of consent that is obtained electronically is not considered written consent unless it is obtained by a method that allows verification of the individual's signature. In other words, saying "yes" by email is rarely considered to be written documentation of consent | | | |
|---|---|---|---|---|
| <b>a.</b> Is written | documentation of consent beir | ng obtained for: | | |
| <b>X</b> None | of the research procedures | → Use the table below to provide justification the 8.5. | nen go to <u>c</u> | question |
| All of | the research procedures | → Do not complete the table; go to question 8.4 | l <u>.b.</u> | |
| Some | of the research procedures | Use the table below to identify the procedure<br>documentation of consent will not be obtaine<br>subjects. | | |
| Adult<br>subject<br>group <sup>1</sup> | | r data/specimen collection (if any) for which<br>NO documentation of consent | provide<br>wri<br>state<br>describ<br>rese | hey be ed with a tten ement bing the earch onal)? |
| Parent/<br>guardian | summary of the research proje | of Parent/ guardian permission. We will provide a ects. Ask parents to check yes/no indicating their to and mail the complete study information. | х | |
| Table footnotes | | | | |

**8.4 Written documentation of consent.** Which of the statements below describe whether documentation of consent will be obtained? NOTE: This question does not apply to screening and recruiting procedures which have already

been addressed in question 4.7.

1. If the answer is the same for all adult groups or all procedures, collapse the answer across the groups and/or procedures.

- **b. Electronic consent signature.** For studies in which documentation of consent will be obtained: will subjects use an electronic method to provide their consent signature?
  - See the <u>GUIDANCE Electronic Informed Consent</u> for information about options (including REDCap e-signature and the DocuSign system) and any associated requirements.
  - FDA-regulated studies must use a system that complies with the FDA's "Part 11" requirements about electronic systems and records. Note that the UW-IT supported DocuSign e-signature system does not meet this requirement.
  - Having subjects check a box at the beginning of an emailed or web-based questionnaire is not considered legally effective documentation of consent.

| X | No | | | |
|---|---|---|---|---|
| | Yes | → If yes | , indicate which methodo | logy will be used. |
| | | | UW ITHS REDCap | |
| | | | Other REDCap<br>installation | → Please name the institutional version you will be using (e.g. Vanderbilt, Univ. of Cincinnati) in the field below and provide a completed <b>SUPPLEMENT Other REDCap</b> Installation with your submission. |
| | | | UW DocuSign | |
| | | | Other | → Please describe in the field below |
| | | b.1 | Is this method legally valid | I in the jurisdiction where the research will occur? |
| | | | NOTE: UW ITHS REDCap a and federal laws regarding | nd UW DocuSign have been vetted for compliance with WA State |

**b.2** Will verification of the subject's identity be obtained if the signature is not personally witnessed by a member of the study team? Note that this is required for FDA-regulated studies.

| No →If no, provide the rationale for why this is not required or necessary to protest subjects or the integrity of the research. Also, what would be the risks to the actual subject if somebody other than the intended signer provides the consistency. | |
|---|---|
| | Yes →If yes, describe how subject identity will be verified, providing a non- technical |
| | description that the reviewer will understand. |
| | b.3 How will the requirement be met to provide a copy of the consent information (consent form) to individuals who provide an e-signature? |
| | The copy can be paper or electronic and may be provided on an electronic storage device or via email. If the electronic consent information uses hyperlinks or other websites or podcasts to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. |
| or who lack f | speaking or -reading adult subjects. Will the research enroll adult subjects who do not speak English luency or literacy in English? If yes, describe the process that will be used to ensure that the oral and written information provided to them during the consent process and throughout the study will be in a language readily understandable to them and (for written materials such as consent forms or questionnaires) at an appropriate reading/comprehension level. |
| | <b>a.</b> <u>Interpretation</u> . Describe how interpretation will be provided, and when. Also, describe the qualifications of the interpreter(s) – for example, background, experience, language proficiency in English and in the other language, certification, other credentials, familiarity with the research-related vocabulary in English and the target language. |
| | <b>b.</b> <u>Translations</u> . Describe how translations will be obtained for all study materials (not just consent forms). Also, describe the method for ensuring that the translations meet the UW IRB's requirement that translated documents will be linguistically accurate, at an appropriate reading level for the participant population, and culturally sensitive for the locale in which they will be used. |

See the <u>GUIDANCE Electronic Informed Consent</u> for information and examples

8.6 Barriers to written documentation of consent. There are many possible barriers to obtaining written documentation of consent. Consider, for example, individuals who are functionally illiterate; do not read English well; or have sensory or motor impairments that may impede the ability to read and sign a consent form. a. Describe the plans (if any) for obtaining written documentation of consent from potential subjects who may have difficulty with the standard documentation process (that is, reading and signing a consent form). Skip this

question if written documentation of consent is not being obtained for any part of the research.

Examples of solutions: Translated consent forms; use of the Short Form consent process; reading the form to the person before they sign it; excluding individuals who cannot read and understand the consent form.

The study permission form follows the same process and is written at the same language level as other documents and permission forms. We will add in the option that the parent can request a call or video conference meetings with the PI and PD for a one-to-one meeting. The PI (UW) or PD (

| | explain the study, read the permission form, pausing after each section and ask if they have questions. Once the permission form is read, the PI/PD will ask them to verbally share their understanding of the program and correct any misunderstanding. After the reading, the PI/PD will ask if their student has their permission to participate, if so the parent may make their mark on the form and a witness approved by the parent will sign the form. |
|---|---|
| | <b>ception</b> . Will information be deliberately withheld, or will false information be provided, to any of the subjects? |
| | e: "Blinding" subjects to their study group/condition/arm is not considered to be deception, but not telling them ahead of e that they will be subject to an intervention or about the purpose of the procedure(s) is deception. |
| X | No |
| | Yes → If yes, describe what information and why. |
| | Example: It may be necessary to deceive subjects about the purpose of the study (describe why). |
| | a. Will subjects be informed beforehand that they will be unaware of or misled regarding the<br>nature or purposes of the research? (Note: this is not necessarily required.) |
| | No<br>Yes |
| | <b>b.</b> Will subjects be debriefed later? (Note: this is not necessarily required.) |
| | No Yes → If yes, describe how and when this will occur. Upload any debriefing materials, including talking points or a script, to <i>Zipline</i> . |
| 3.8 Cog | nitively impaired adults, and other adults unable to consent. Will such individuals be included in the |

( research?

Examples: individuals with Traumatic Brain Injury (TBI) or dementia; individuals who are unconscious, or who are significantly intoxicated.

| Х | No | → If no, go to question <b>8.9</b> . |
|---|-----|---------------------------------------------------|
| | Yes | ightarrow If yes, answer the following questions. |

| b. Capacity for consent / decision making capacity. Describe the process that will be used to determine whether a cognitively impaired individual is capable of consent decision making with respect to the research protocol and setting. |
|---|
| b.1. If there will be repeated interactions with the impaired subjects over a time period when cognitive capacity could increase or diminish, also describe how (if at all) decision-making capacity will be re-assessed and (if appropriate) consent obtained during that time. |
| c. <u>Permission (surrogate consent)</u> . If the research will include adults who cannot consent for<br>themselves, describe the process for obtaining permission ("surrogate consent") from a legally<br>authorized representative (LAR). |
| For research conducted in Washington State, see the <b>GUIDANCE Legally Authorized Representative</b> to learn which individuals meet the state definition of "legally authorized representative". |
| d. <u>Assent</u> . Describe whether assent will be required of all, some, or none of the subjects. If some, indicate which subjects will be required to assent and which will not (and why not). Describe any process that will be used to obtain and document assent from the subjects. |
| e. <u>Dissent or resistance</u> . Describe how a subject's objection or resistance to participation (including non-verbal) during the research will be identified, and what will occur in response. |
| <b>8.9 Research use of human fetal tissue obtained from elective abortion.</b> Federal and UW Policy specify some requirements for the consent process. If you are conducting this type of research, check the boxes to confirm these requirements will be followed. |
| Informed consent for the donation of fetal tissue for research use will be obtained by someone other than |
| the person who obtained the informed consent for abortion. Informed consent for the donation of fetal tissue for research use will be obtained after the informed consent for abortion. |
| Participation in the research will not affect the method of abortion. |
| No enticements, benefits, or financial incentives will be used at any level of the process to incentivize |
| abortion or the donation of human fetal tissue. The informed consent form for the donation of fetal tissue for use in research will be signed by both the |
| Document Date & Version Researcher Date & Version |
| 01/21/2021 10/04/2022 |

**a.** Rationale. Provide the rationale for including this population.

woman and the person who obtains the informed consent.

- **8.10 Consent-related materials**. Upload to *Zipline* all consent scripts/talking points, consent forms, debriefing statements, Information Statements, Short Form consent forms, parental permission forms, and any other consent-related materials that will be used. Materials that will be used by a specific site should be uploaded to that site's **Local Site Documents** page.
  - <u>Translations must be submitted and approved before they can be used</u>. However, we strongly encourage you to wait to provide them until the IRB has approved the English versions.
  - <u>Combination forms</u>: It may be appropriate to combine parental permission with consent, if parents are subjects as well as providing permission for the participation of their children. Similarly, a consent form may be appropriately considered an assent form for older children.
  - For materials that cannot be uploaded: upload screenshots or written descriptions that are sufficient to enable the IRB to understand the types of data that will be collected and the nature of the experience for the participant. URLs (website addresses) may also be provided, or written descriptions of websites. Examples of materials that usually cannot be uploaded: mobile apps; computer-administered test; licensed and restricted standardized tests.

## 9 PRIVACY AND CONFIDENTIALITY

**9.1 Privacy protections.** Describe the steps that will be taken, if any, to address possible privacy concerns of subjects and potential subjects.

Privacy refers to the sense of being in control of access that others have to ourselves. This can be an issue with respect to recruiting, consenting, sensitivity of the data being collected, and the method of data collection. Examples:

- Many subjects will feel a violation of privacy if they receive a letter asking them to participate in a study because they
  have \_\_\_\_ medical condition, when their name, contact information, and medical condition were drawn from medical
  records without their consent. Example: the IRB expects that "cold call" recruitment letters will inform the subject
  about how their information was obtained.
- Recruiting subjects immediately prior to a sensitive or invasive procedure (e.g., in an outpatient surgery waiting room) will feel like an invasion of privacy to some individuals.
- Asking subjects about sensitive topics (e.g. details about sexual behavior) may feel like an invasion of privacy to some individuals.

If a participant chooses to participate in the Digital Storytelling portion of the program, they will be trained in how to design and develop their own short story using digital cameras, digital video cameras, and digital audio recorders. There is likely to be little to no discomfort in sharing their story since they will be in charge of deciding what information they want to share. Photos collected during the activities and throughout the program are theirs to keep and not used for research purposes.

We will provide the following information in both the permission form and a simplified version in the assent form:

Participants may be worried about people finding out what they say in these assessments or activities. There is a risk of loss of confidentiality (i.e., someone outside the study finding out personal information about a participant). We will take several steps to protect participants from these risks, and these protections are described here:

The information given to us will be used for research purposes only and will be kept private. Names and other identifiers will not be put directly on the participant's survey response. Instead, the data will be given an ID number, and the ID number will be linked to names and identifiers on a list that will be kept separate from the

data in a secure location. Therefore, it would be difficult for anybody outside the research team to identify any person's answers.

We will inform participants that there are exceptions to our ability to keep what we learn private. If they tell us that a child or elder is being abused, we may need to report it to authorities. Also, we may need to call authorities if we think they are at risk of hurting yourself or someone else. Government or university staff sometimes review studies such as this one to make sure they are being done safely and legally. If a review of this study takes place, someone may look at participant records. The reviewers will protect participant privacy and study records will not be used to put participants at legal risk of harm.

We will receive community approval before publishing or presenting any of the results. In any sort of report we might publish, we will not include any information that will make it possible to identify a person. If they would like to see a copy of the final report once the study is finished, they can contact Dr. Teresa Evans-Campbell (206) 543-6075 tecamp@uw.edu at the University of Washington Indigenous Wellness Research Institute.

| 9.2 | Identification of individuals in publications and presentations. Will potentially identifiable information about |
|---|---|
| | subjects be used in publications and presentations, or is it possible that individual identities could be inferred from |
| | what is planned to be published or presented? |

| X | No | | | |
|---|---|---|---|---|
| | Yes | $\rightarrow$ If ye | s, will su | bject consent be obtained for this use? |
| | | | Yes | |
| | | | No | → If no, describe the steps that will be taken to protect subjects (or small groups of |
| | | | = | subjects) from being identifiable. |

- (9.3) State mandatory reporting. Each state has reporting laws that require some types of individuals to report some kinds of abuse, and medical conditions that are under public health surveillance. These include:
  - Child abuse
  - Abuse, abandonment, neglect, or financial exploitation of a vulnerable adult
  - Sexual assault
  - Serious physical assault
  - Medical conditions subject to mandatory reporting (notification) for public health surveillance

Are you or a member of the research team likely to learn of any of the above events or circumstances while conducting the research **AND** feel obligated to report it to state authorities?

No X Yes

→ If yes, the UW IRB expects subjects to be informed of this possibility in the consent form or during the consent process, unless you provide a rationale for not doing so:

We will provide this information in the permission and assent form

**9.4 Retention of identifiers and data.** Check the box below to indicate assurance that any identifiers (or links between identifiers and data/specimens) and data that are part of the research records will not be destroyed until after the end of the applicable records retention requirements (e.g. Washington State; funding agency or sponsor; Food and Drug Administration). If it is important to say something about destruction of identifiers (or links to identifiers) in the consent form, state something like "the link between your identifier and the research data will be destroyed after the records retention period required by state and/or federal law."

This question can be left blank for conversion applications (existing paper applications that are being "converted" into a Zipline application.)

See the "Research Data" sections of the following website for UW Records management for the Washington State research rectords retention schedules that apply in general to the UW (not involving UW Medicine data): <a href="http://f2.washington.edu/fm/recmgt/gs/research?title=R">http://f2.washington.edu/fm/recmgt/gs/research?title=R</a>

See the "Research Records and Data" information in Section 8 of this document for the retention schedules for UW Medicine Records: <a href="https://www.uwmedicine.org/recordsmanagementuwm-records-retention-schedule.pdf">https://www.uwmedicine.org/recordsmanagementuwm-records-retention-schedule.pdf</a>

X Confirm

**9.5 Certificates of Confidentiality**. Will a federal Certificate of Confidentiality be obtained for the research data? *NOTE: Answer "No" if the study is funded by NIH or the CDC, because all NIH-funded and CDC-funded studies automatically have a Certificate.* 

X No Yes

- (9.6) Data and specimen security protections. Identify the data classifications and the security protections that will be provided for all sites where data will be collected, transmitted, or stored, referring to the GUIDANCE Data and Security Protections for the minimum requirements for each data classification level. It is not possible to answer this question without reading this document. Data security protections should not conflict with records retention requirements.
  - **a.** Which level of protections will be applied to the data and specimens? If more than one level will be used, describe which level will apply to which data and which specimens and at which sites.

Level 4: Would likely cause serious harm to individuals if disclosed

**b.** Use this space to provide additional information, details, or to describe protections that do not fit into one of the levels. If there are any protections within the level listed in 9.6.a which will *not* be followed, list those here, including identifying the sites where this exception will apply.

We intend to comply with all of level 4 protections

## **10 RISK / BENEFIT ASSESSMENT**

- **10.1** Anticipated risks. Describe the <u>reasonably foreseeable</u> risks of harm, discomforts, and hazards to the subjects and others of the research procedures. For each harm, discomfort, or hazard:
  - Describe the magnitude, probability, duration, and/or reversibility of the harm, discomfort, or hazard, AND
  - Describe how the risks will be reduced or managed. Do not describe data security protections here, these are already described in Question 9.6.
  - Consider possible physical, psychological, social, legal, and economic harms, including possible negative effects on financial standing, employability, insurability, educational advancement or reputation. For example, a breach of confidentiality might have these effects.
  - Examples of "others": embryo, fetus, or nursing child; family members; a specific group.
  - Ensure applicable risk information from any Investigator Brochures, Drug Package Inserts, and/or Device Manuals is included in your description.
  - Do not include the risks of non-research procedures that are already being performed.
  - If the study design specifies that subjects will be assigned to a specific condition or intervention, then the condition or intervention is a research procedure even if it is a standard of care.
  - Examples of mitigation strategies: inclusion/exclusion criteria; applying appropriate data security measures to prevent unauthorized access to individually identifiable data; coding data; taking blood samples to monitor something that indicates drug toxicity.
  - As with all questions on this application, you may refer to uploaded documents.

Participants will be asked about thoughts, feelings, and personal difficulties that may be private and feel sensitive. They may feel embarrassed or anxious if they choose to disclose personal information. They will be asked about trauma exposure, and health behaviors and about potentially illegal behaviors such as substance use. These questions may make them feel uncomfortable, bring back stressful or upsetting memories or seem intrusive. If they experience an increase in emotional distress related to their participation in the project, they are asked to let study staff know so that we can provide appropriate support.

They may also worry about people finding out what they say in these assessments or activities. There is a risk of loss of confidentiality (i.e., someone outside the study finding out personal information about them). We have taken several steps to protect them from these risks as noted in 9.1 above.

During the optional outdoor activities, they may feel environmentally-based discomfort related to heat or rain exposure, limited bathroom access, walking on some unpaved roads, roads with hills, curves, or construction work, as well as exposure to insects such as ticks or mosquitos, wildlife such as snakes, and flora or fauna such as poison oak or ivy. At any time, if they need a break, vehicles will be in close proximity for easy access, extra hydration, and rest and vehicles to transport more significant injuries to appropriate medical resources. As a student, they can access the IHS health clinic services on campus free of charge.

Reproductive risks. Are there any risks of the study procedures to men and women (who are subjects, or partner of subjects) related to pregnancy, fertility, lactation or effects on a fetus or neonate?

Examples: direct teratogenic effects; possible germline effects; effects on fertility; effects on a woman's ability to continue a pregnancy; effects on future pregnancies.

| X | No | → If no go to question 10.3 |
|---|---|---|
| | Yes | → If yes, answer the following questions: |
| | | a. Risks. Describe the magnitude, probability, duration and/or reversibility of the risks. |

**b. Steps to minimize risk**. Describe the specific steps that will be taken to minimize the magnitude, probability, or duration of these risks.

Examples: inform the subjects about the risks and how to minimize them; require a pregnancy test before and during the study; require subjects to use contraception; advise subjects about banking of sperm and ova.

If the use of contraception will be required: describe the allowable methods and the time period when contraception must be used.

c. Pregnancy. Describe what will be done if a subject (or a subject's partner) becomes pregnant

For example; will subjects be required to immediately notify study staff, so that the study procedures can be discontinue or modified, or for a discussion of risks, and/or referrals or counseling?

- **MRI risk management.** A rare but serious adverse reaction called nephrogenic systemic fibrosis (NSF) has been observed in individuals with kidney disease who received gadolinium-based contrast agents (GBCAs) for the scans. Also, a few healthy individuals have a severe allergic reaction to GBCAs.
  - a. Use of gadolinium. Will any of the MRI scans involve the use of a gadolinium-based contrast agent (GBCA?)

X No Yes

→ If yes, which agents will be used? Check all that apply.

| Brand Name | Generic Name | Chemical Structure |
|----------------------|--------------------------|--------------------|
| Dotarem | Gadoterate meglumine | Macrocylic |
| Eovist / Primovist | Gadoxetate disodium | Linear |
| Gadavist | Gadobutro | Macrocyclic |
| Magnevist | Gadpentetate dimeglumine | Linear |
| MultiHance | Gadobenate dimeglumine | Linear |
| Omniscan | Gadodiamide | Linear |
| OptiMARK | Gadoversetamide | Linear |
| ProHance | Gadoteridol | Macrocyclic |
| Other, provide name: | | |

| | significantly longer time than previously recognized, especially for linear GBCAs. The health-related risks of this longer retention are not yet clearly established. However, the UW IRB expects researchers to provide a compelling justification for using a linear GBCA instead of a macrocyclic GBCA, to manage the risks associated with GBCAs. |
|---|---|
| | Describe why it is important to use a GBCA with the MRI scan(s). Describe the dose that will be used and (if it is more than the standard clinical dose recommended by the manufacturer) why it is necessary to use a higher dose. If a linear GBCA will be used, explain why a macrocyclic GBCA cannot be used. |
| 2.) | Information for subjects. Confirm by checking this box that subjects will be provided with the FDA-approved Patient Medication Guide for the GBCA being used in the research or that the same information will be inserted into the consent form. Confirmed |
| | ose of GBCA; (2) prepare it for injection; (3) insert and remove the IV catheter; (4) (5) monitor for any adverse effects of the GCBA? Also, what are the qualifications dual(s)? |
| <ul><li>c. Describe how the renal fun<br/>be used to exclude subject</li></ul> | ction of subjects will be assessed prior to MRI scans and how that information will s at risk for NSF. |
| • | andling a severe allergic reaction to the GBCA or any other medical ne MRI scan, including who will be responsible for which actions. |
| event/emergency during t | , |
| event/emergency during t | |
| | re any research procedures that may have risks that are currently unforeseeable? |
| 10.4 Unforeseeable risks. Are the | |
| Unforeseeable risks. Are then Example: using a drug that hasn No | re any research procedures that may have risks that are currently unforeseeable? It been used before in this subject population. |
| Unforeseeable risks. Are then Example: using a drug that hasn No | re any research procedures that may have risks that are currently unforeseeable? |

| Yes → If yes, check all the boxes that apply. |
|---|
| Administration of any drug for research purposes |
| Inserting an intra-venous (central or peripheral) or intra-arterial line for research purposes |
| Obtaining samples of blood, urine, bone marrow or cerebrospinal fluid for research purposes |
| Obtaining a research sample from tissue or organs that would not otherwise be removed during surgery |
| Administration of a radio-isotope for research purposes** |
| Implantation of an experimental device |
| Other manipulations or procedures performed solely for research purposes (e.g., experimental liver dialysis, experimental brain stimulation) |
| If any of the boxes are checked: Provide the name and institutional affiliation of a physician anesthesiologist who is a member of the research team or who will serve as a safety consultant about the interactions between the research procedures and the general or regional anesthesia of the subject-patients. If the procedures will be performed at a UW Medicine facility or affiliate, the anesthesiologist must be a UW faculty member, and the Vice Chair of Clinical Research in the UW Department of Anesthesiology and Pain Medicine must be consulted in advance for feasibility, safety and billing. |
| ** If the box about radio-isotopes is checked: the study team is responsible for informing in advance all appropriate clinical personnel (e.g., nurses, technicians, anesthesiologists, surgeons) about the administration and use of the radio-isotope, to ensure that any personal safety issues (e.g., pregnancy) can be appropriately addressed. This is a condition of IRB approval. |
| 6 Data and Safety Monitoring. A Data and Safety Monitoring Plan (DSMP) is required for clinical trials (as defined by NIH). If required for this research, or if there is a DSMP for the research regardless of whether it is required, upload the DSMP to <i>Zipline</i> . If it is embedded in another document being uploading (for example, a Study Protocol) use the text box below to name the document that has the DSMP. Alternatively, provide a description of the DSMP in the text box below. |
| Attached |
| 7 Un-blinding. If this is a double-blinded or single-blinded study in which the participant and/or relevant study team members do not know the group to which the participant is assigned: describe the circumstances under which un-blinding would be necessary, and to whom the un-blinded information would be provided. |
| no |

**10.8 Withdrawal of participants.** If applicable, describe the anticipated circumstances under which participants will be withdrawn from the research without their consent. Also, describe any procedures for orderly withdrawal of a participant, regardless of the reason, including whether it will involve partial withdrawal from procedures and any intervention but continued data collection or long-term follow-up.

n/a

Anticipated direct benefits to participants. If there are any direct research-related benefits that some or all individual participants are likely to experience from taking part in the research, describe them below:

Do not include benefits to society or others, and do not include subject payment (if any). Examples: medical benefits such as laboratory tests (if subjects receive the results); psychological resources made available to participants; training or education that is provided.

Participants may benefit by learning more about themselves through participation in the study, learning about how to make healthy behavioral changes, learning youth leadership skills and learning digital storytelling skills, or going on a field trip.

They may also feel good about helping an effort that is aimed at improving the health and wellness of Native American youth across the country.

## (10.10) Return of individual research results.

In this section, provide your plans for the return of individual results. An "individual research result" is any information collected, generated or discovered in the course of a research study that is linked to the identity of a research participant. These may be results from screening procedures, results that are actively sought for purposes of the study, results that are discovered unintentionally, or after analysis of the collected data and/or results has been completed.

See the <u>GUIDANCE Return of Individual Results</u> for information about results that should and should not be returned, validity of results, the Clinical Laboratory Improvement Amendment (CLIA), consent requirements and communicating results.

a. Is it anticipated that the research will produce any individual research results that are clinically actionable?

"Clinically actionable" means that there are established therapeutic or preventive interventions or other available actions that have the potential to change the clinical course of the disease/condition, or lead to an improved health outcome.

In general, every effort should be made to offer results that are clinically actionable, valid and pose life-threatening or severe health consequences if not treated or addressed quickly. Other clinically actionable results should be offered if this can be accomplished without compromising the research.

X No Yes

→ If yes, answer the following questions (a.1-a.3).

**a.1.** Describe the clinically actionable results that are anticipated and explain which results, if any, could be urgent (i.e. because they pose life-threatening or severe health consequences if not treated or addressed quickly).

Examples of urgent results include very high calcium levels, highly elevated liver function test results, positive results for reportable STDs.

**a.2.** Explain which of these results will be offered to subjects.

| <b>10.11 Co</b> | e. Describe any plans to share results with family members (e.g. in the event a subject becomes incapacitated or deceased). f. Check the box to indicate that any plans for return of individual research results have been described in the consent document. If there are no plans to provide results to participants, this should be stated in the consent form. See the GUIDANCE Return of Individual Results for information about consent requirements. Confirmed mmercial products or patents. Is it possible that a commercial product or patent could result from this addy? No Yes If yes, describe whether subjects might receive any remuneration/compensation and, if yes, how the amount will be determined. |
|---|---|
| <b>10.11 Co</b> | e. Describe any plans to share results with family members (e.g. in the event a subject becomes incapacitated or deceased). f. Check the box to indicate that any plans for return of individual research results have been described in the consent document. If there are no plans to provide results to participants, this should be stated in the consent form. See the GUIDANCE Return of Individual Results for information about consent requirements. Confirmed mmercial products or patents. Is it possible that a commercial product or patent could result from this ady? No |
| 10.11 Co | <ul> <li>e. Describe any plans to share results with family members (e.g. in the event a subject becomes incapacitated or deceased).</li> <li>f. Check the box to indicate that any plans for return of individual research results have been described in the consent document. If there are no plans to provide results to participants, this should be stated in the consent form.</li> <li>See the GUIDANCE Return of Individual Results for information about consent requirements.</li> <li>Confirmed</li> <li>mmercial products or patents. Is it possible that a commercial product or patent could result from this</li> </ul> |
| | e. Describe any plans to share results with family members (e.g. in the event a subject becomes incapacitated or deceased). f. Check the box to indicate that any plans for return of individual research results have been described in the consent document. If there are no plans to provide results to participants, this should be stated in the consent form. See the GUIDANCE Return of Individual Results for information about consent requirements. Confirmed |
| | <ul> <li>e. Describe any plans to share results with family members (e.g. in the event a subject becomes incapacitated or deceased).</li> <li>f. Check the box to indicate that any plans for return of individual research results have been described in the consent document. If there are no plans to provide results to participants, this should be stated in the consent form.</li> </ul> |
| | <ul> <li>e. Describe any plans to share results with family members (e.g. in the event a subject becomes incapacitated or deceased).</li> <li>f. Check the box to indicate that any plans for return of individual research results have been described in the consent document. If there are no plans to provide results to participants, this should be stated in the</li> </ul> |
| | <ul> <li>Describe any plans to share results with family members (e.g. in the event a subject becomes incapacitated or deceased).</li> </ul> |
| | e. Describe any plans to share results with family members (e.g. in the event a subject becomes |
| | e. Describe any plans to share results with family members (e.g. in the event a subject becomes |
| | useu. |
| | communicate the result (if different), the circumstances, timing, and communication methods that will be used. |
| | <b>d</b> . Describe the process for communicating results to subjects and facilitating understanding of the results. In the description, include who will approach the participant with regard to the offer of results, who will be appropriate the result (if different), the circumstance of timing and communication methods that will be |
| | The IRB will consider evidence of validity such as studies demonstrating diagnostic, prognostic, or predictive value, use of confirmatory testing, and quality management systems. |
| | c. Describe the validity and reliability of any results that will be offered to subjects. |
| | Yes → If yes, explain which results will be offered to subjects and provide the rationale for offering these results. |
| | Examples: non-actionable genetic results, clinical tests in the normal range, experimental and/or uncertain results. No |
| | <b>b</b> . Is there a plan for offering subjects any results that are <u>not</u> clinically actionable? |
| | <ul> <li>There are insufficient resources to communicate the results effectively and appropriately</li> <li>Knowledge of the result could cause psychosocial harm to subjects</li> </ul> |
| | <ul> <li>There are serious questions regarding validity or reliability</li> <li>Returning the results has the potential to cause bias</li> </ul> |

**a.3.** Explain which results will <u>not</u> be offered to subjects and provide the rationale for not

offering these results.

## 11 ECONOMIC BURDEN TO PARTICIPANTS

**11.1 Financial responsibility for research-related injuries.** Answer this question only if the lead researcher is <u>not</u> a UW student, staff member, or faculty member whose primary paid appointment is at the UW.

For each institution involved in conducting the research: Describe who will be financially responsible for research-related injuries experienced by subjects, and any limitations. Describe the process (if any) by which participants may obtain treatment/compensation.

N/A

**11.2 Costs to subjects**. Describe any research-related costs for which subjects and/or their health insurance may be responsible (examples might include: CT scan required for research eligibility screening; co-pays; surgical costs when a subject is randomized to a specific procedure; cost of a device; travel and parking expenses that will not be reimbursed).

N/A

## **12 RESOURCES**

- **12.1** Faculty Advisor. (For researchers who are students, residents, fellows, or post-docs.) Provide the following information about the faculty advisor.
  - Advisor's name
  - Your relationship with your advisor (for example: graduate advisor; course instructor)
  - Your plans for communication/consultation with your advisor about progress, problems, and changes.

N/A

**12.2 UW Principal Investigator Qualifications.** Upload a current or recent Curriculum Vitae (CV), Biosketch (as provided to federal funding agencies), or similar document to the Local Site Documents page in Zipline. The purpose of this is to address the PI's qualifications to conduct the proposed research (education, experience, training, certifications, etc.).

For help with creating a CV, see <a href="http://adai.uw.edu/grants/nsf\_biosketch\_template.pdf">https://education.uwmedicine.org/student-affairs/career-advising/year-4/residency-applications/curriculum-vitae/</a>

- X The CV will be uploaded.
- 12.3 UW Study team qualifications. Describe the qualifications and/or training for each <u>UW</u> study team member to fulfill their role on the study and perform study procedures. (You may be asked about non-UW study team members during the review; they should not be described here.) You may list these individuals by name, however if you list an individual by name, you will need to modify this application if that individual is replaced. Alternatively, you can describe study <u>roles</u> and the qualifications and training the PI or study leadership will require for any individual who might fill that role. The IRB will use this information to assess whether risks to subjects are minimized because study activities are being conducted by properly qualified and trained individuals.

Describe: The role (or name of person), the study activities they will perform, and the qualifications or training that are relevant to performing those study activities.

### **Examples:**

<u>Research Study Coordinator:</u> Obtain consent, administer surveys, blood draw. Will have previous experience coordinating clinical research and be a certified phlebotomist in WA.

<u>Undergraduate Research Assistant:</u> Obtain consent, perform all study procedures. Will have had coursework in research methods, complete an orientation to human subjects protections given by the department, and will receive training from the PI or the graduate student project lead on obtaining consent and debriefing subjects. <u>Acupuncturist:</u> Perform acupuncture procedures and administer surveys. Must be licensed with WA State DoH and complete training in administering research surveys given by the project director, an experienced survey researcher.

<u>Co-Investigator:</u> Supervise MRI and CT scan procedures and data interpretation, obtain consent. MD, specialty in interventional radiology and body imaging. 5-years clinical research experience.

Study coordinator: manage the day to day field operations. Will have a master degree and 2+ years experience managing clinical trials.

Co-Investigators (3):

- 1. Provide expertise in implementing behavioral health clinical trials among Native Americans 10+ year experience.
- 2. Expertise in training and supervising counselors in motivational interviewing (MI) 10 year plus experince
- 3. Conducting statistical analysis and ensuring data quality. 5 year plus experience

| <b>12.4 Study team training and communication</b> . Describe how it will be ensured that each study team member is | |
|---|---|
| | adequately trained and informed about the research procedures and requirements (including any changes) as |
| | well as their research-related duties and functions. |

| There | is | no | study | team. |
|-------|----|----|-------|--------|
| | | | Juan | ccaiii |

All staff will hold certificates in human subject training; investigators will have certificate in Good Clinical Practice; PI will meet with the Research coordinator and site staff 2-3 times a month or more often as needed.

# 13 OTHER APPROVALS, PERMISSIONS, and REGULATORY ISSUES

Approvals and permissions. Identify any other approvals or permissions that will be obtained. For example: from a school, external site/organization, funding agency, employee union, UW Medicine clinical unit.

Do not attach the approvals and permissions unless requested by the IRB.

Principal letter of support/approval

**13.2 Financial Conflict of Interest.** Does any UW member of the team have ownership or other Significant Financial Interest (SFI) with this research as defined by UW policy GIM 10?



| Yes | → If yes, has the proposed res | e Office of Research made a determination regarding this SFI as it pertains to the search? |
|---|---|---|
| | No | → If no, contact the Office of Research (206.616.0804, <a href="mailto:research@uw.edu">research@uw.edu</a> ) for guidance on how to obtain the determination |
| | Yes | → If yes, upload the Conflict Management Plan for every UW team member who has a FCOI with respect to the research, to <i>Zipline</i> . If it is not yet available, use the text box to describe whether the Significant Financial Interest has been disclosed already to the UW Office of Research and include the FIDS Disclosure ID if available. |

(13.3) UW ITHS COVID review. Confirm by checking the box that you will obtain this additional review if it is applicable to your research (see "Proposal Eligibility" at this link <a href="https://www.iths.org/iths-covid-19-research-resources/covid-19-research-portal/">https://www.iths.org/iths-covid-19-research-resources/covid-19-research-portal/</a>).

Confirmed